# 1.0 Title Page

# **Statistical Analysis Plan**

# **Study M15-925**

A Phase 3, Randomized, Active-Controlled, Double-Blind Study Comparing Upadacitinib to Abatacept in Subjects with Moderately to Severely Active Rheumatoid Arthritis with Inadequate Response or Intolerance to Biologic DMARDs (bDMARDs) on Stable Conventional Synthetic Disease Modifying Anti-Rheumatic Drugs (csDMARDs)

**Date: 17 Dec 2020** 

Version 2.0

| 2.0 | Table of Contents | |
|---|---|---|
| 1.0 | Title Page | 1 |
| 2.0 | Table of Contents | <mark>2</mark> |
| 3.0 | Introduction | <mark>7</mark> |
| 4.0 | Study Objectives, Design and Procedures | <mark>7</mark> |
| 4.1 | Study Objectives | 7 |
| 4.2 | Overall Study Design and Plan | 7 |
| 4.3 | Study Design History | 11 |
| 4.4 | Sample Size | 12 |
| 4.5 | Interim Analysis and Date Base Lock | 13 |
| 4.6 | Data Monitoring Committee (DMC) Activities | 13 |
| 5.0 | Analysis Populations and Analysis Windows | 13 |
| 5.1 | Analysis Populations | 13 |
| 5.2 | Analysis Windows | 14 |
| 6.0 | Demographics, Baseline Characteristics, Medical History, and Previous/Concomitant Medications | 17 |
| 6.1 | Demographics and Baseline Characteristics | 17 |
| 6.2 | Medical History | 20 |
| 6.3 | Prior Treatment and Concomitant Medications | 21 |
| 6.4 | Protocol Deviations | 21 |
| 7.0 | Patient Disposition | 22 |
| 8.0 | Study Drug Exposure and Compliance | 23 |
| 8.1 | Study Drug Exposure | 23 |
| 8.2 | Compliance | 24 |
| 9.0 | Efficacy Analysis | 25 |
| 9.1 | General Considerations | 25 |
| 9.1.1 | Efficacy Analysis at Different Phases of the Study | 25 |
| 9.1.2 | Definition of Missing Data Imputation | 25 |
| 9.2 | Efficacy Analysis for Period 1 | 27 |
| 9.2.1 | Primary Efficacy Analysis | 27 |
| 9.2.2 | Sensitivity Analysis of Primary Efficacy Variables | 28 |
| 9.2.3 | Key Secondary Efficacy Analyses | 28 |

| 9.2.4 | Exploratory Efficacy Analyses | 29 |
|---|---|---|
| 9.2.5 | Handling of Multiplicity | 30 |
| 9.2.6 | Efficacy Subgroup Analysis | 30 |
| 9.3 | Long-Term Efficacy Analysis | 31 |
| 9.4 | Efficacy Variables Definitions and Conventions | 32 |
| 9.4.1 | ACR Criteria | 32 |
| 9.4.2 | Joint Evaluation | 35 |
| 9.4.3 | Patient's Global Assessment of Disease Activity Visual Analog<br>Scale (VAS) | 36 |
| 9.4.4 | Physician's Global Assessment of Disease Activity Visual Analog Scale (VAS) | 37 |
| 9.4.5 | Patient's Global Assessment of Pain | 37 |
| 9.4.6 | Disease Activity Score (DAS28) | 37 |
| 9.4.7 | Simplified Disease Activity Index (SDAI) | 38 |
| 9.4.8 | Clinical Disease Activity Index (CDAI) | 38 |
| 9.4.9 | Clinical Remission (CR) and Low Disease Activity (LDA) | 39 |
| 9.4.10 | ACR/EULAR Boolean Remission | 39 |
| 9.4.11 | Disability Index of Health Assessment Questionnaire (HAQ DI) | 39 |
| 9.4.12 | EuroQoL-5D (EQ-5D-5L) | 40 |
| 9.4.13 | Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | 40 |
| 9.4.14 | Form SF-36v2 | 41 |
| 9.4.15 | Work Productivity and Activity Impairment (WPAI) | 41 |
| 9.4.16 | Systemic Corticosteroid Dose | 42 |
| 10.0 | Safety Analysis | 42 |
| 10.1 | General Considerations | 42 |
| 10.2 | Analysis of Adverse Events | 43 |
| 10.2.1 | Analysis of Adverse Events for Period 1 | 44 |
| 10.2.1.1 | Adverse Events Overview | 44 |
| 10.2.1.2 | Adverse Events by System Organ Class and Preferred Term | 45 |
| 10.2.1.3 | TEAEs by Maximum Severity | 45 |
| 10.2.1.4 | TEAEs by Relationship | 46 |

| 10.2.1.5 | Frequent (≥ 2%) Adverse Events and Reasonably Possibly | |
|---|---|---|
| 10.2.1.3 | Related Adverse Events by System Organ Class and Preferred | |
| | Term | 46 |
| 10.2.1.6 | Adverse Events of Special Interest | 46 |
| 10.2.2 | Analysis of Long-Term Adverse Event Rates | 48 |
| 10.2.2.1 | Overview of Adverse Events Rates per 100 Patient-Years of Study Drug Exposure | |
| 10.2.2.2 | Adverse Events Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT | 50 |
| 10.2.2.3 | Adverse Events of Special Interest Rates per 100 Patient Years of Study Drug Exposure | 50 |
| 10.2.2.4 | Listing of Serious Adverse Events (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation | 50 |
| 10.3 | Analysis of Laboratory Data | 50 |
| 10.3.1 | Variables and Units | 50 |
| 10.3.2 | Analysis of Laboratory Data for Period 1 | 52 |
| 10.3.2.1 | Assessment of Mean Change from Baseline and Percentage Change from Baseline in Clinical Laboratory Variables | 53 |
| 10.3.2.2 | Assessment of Shift from Baseline in Clinical Laboratory Variables | 53 |
| 10.3.2.3 | Assessment of Potentially Clinical Significant Laboratory Values | 54 |
| 10.3.2.4 | Assessment of Liver Elevations | 54 |
| 10.3.3 | Analysis of Long-Term Laboratory Data | 55 |
| 10.3.3.1 | Assessment of Mean Change from Baseline and Percentage Change from Baseline in Clinical Laboratory Variables | 55 |
| 10.3.3.2 | Assessment of Potentially Clinically Significant Laboratory Values | 55 |
| 10.3.3.3 | Assessment of Liver Elevations | 56 |
| 10.4 | Analysis of Vital Signs | 56 |
| 10.4.1 | Variables and Criteria Defining Abnormality | 56 |
| 10.4.2 | Analysis of Vital Sign for Period 1 | 57 |
| 10.4.3 | Analysis of Long-Term Vital Sign | 57 |
| 11.0 | Summary of Changes | 58 |

| 11.1 | Summary of Changes between the Previous Version and the Current Version | 58 |
|---|---|---|
| 12.0 | Version History | |
| 13.0 | Appendix | |
| List of Tab | les | |
| Table 1. | Analysis Windows for Efficacy Analysis for Period 1 (for ACR Components and Morning Stiffness) and Safety Analysis for Period 1 (for Labs and Vital Signs) | 15 |
| Table 2. | Analysis Windows for Efficacy Analysis for Period 1 (for EQ 5D 5L and SF-36) | |
| Table 3. | Analysis Windows for Efficacy Analysis for Period 1 (for FACIT-F) | |
| Table 4. | Analysis Windows for Efficacy Analysis for Period 1 (for WPAI) | 16 |
| Table 5. | Insert Table Title Here | 31 |
| Table 6. | Anatomical Joints Assessed for Calculation of Tender and Swollen Joint Counts (TJC68 and SJC66) | 36 |
| Table 7. | Anatomical Joints for DAS28 (CRP) Calculation | 38 |
| Table 8. | AESI for Upadacitinib with SMQs/CMQs/PTs Searches | 47 |
| Table 9. | List of Laboratory Variables | 51 |
| Table 10. | Criteria for Potentially Clinically Significant Vital Sign Findings | 57 |
| Table 11. | SAP Version History Summary | 59 |
| List of Fig | ures | |
| Figure 1. | Period 1 Study Design | 10 |
| Figure 2. | Period 2 Study Design | 11 |
| List of App | pendices | |
| Appendix A. | Statistical Analysis for the 30 mg Cohort | 60 |
| Appendix B. | Statistical Analysis to Account for Impact of COVID-19 Pandemic | 63 |



| Appendix C. | OMERACT Criteria | 65 |
|-------------|------------------|----|
| 1 1 | | |



### 3.0 Introduction

This statistical analysis plan (SAP) describes the statistical analyses to be completed by the Data and Statistical Science Department for Upadacitinib Study M15-925. It provides details to further elaborate statistical methods as outlined in the protocol. Pharmacokinetic and biomarker analyses will be performed separately and the corresponding analysis plan is documented separately.

Unless noted otherwise, all analyses will be performed using SAS version 9.2 or later (SAS Institute Inc., Cary, NC 27513) under the UNIX operating system.

# 4.0 Study Objectives, Design and Procedures

# 4.1 Study Objectives

#### Period 1

To compare the safety and efficacy of upadacitinib 15 mg once daily (QD) versus abatacept intravenous (IV) for the treatment of signs and symptoms of rheumatoid arthritis (RA) in bDMARD-inadequate response (bDMARD-IR) or bDMARD-intolerant subjects on stable conventional synthetic DMARDs with moderately to severely active RA.

#### Period 2

To evaluate the long-term safety, tolerability, and efficacy of Upadacitinib 15 mg QD in subjects with RA who have completed Period 1.

# 4.2 Overall Study Design and Plan

This is a Phase 3, multicenter study that includes two periods. Period 1 is a 24-week randomized, double-blind, parallel-group, active-controlled treatment period designed to compare the safety and efficacy of upadacitinib 15 mg QD versus abatacept IV for the treatment of signs and symptoms of subjects with moderately to severely active RA who have an inadequate response to or intolerance to bDMARD therapies other than abatacept



and are currently on a stable dose of csDMARDs. Period 2 is an open-label extension to evaluate the long-term safety, tolerability, and efficacy of upadacitinib 15 mg QD in subjects with RA who have completed Period 1. Starting with Amendment 5, all subjects will receive open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 mg QD.

The study is designed to enroll approximately 550 subjects at approximately 200 study centers worldwide to meet scientific and regulatory objectives without enrolling an undue number of subjects in alignment with ethical considerations. Therefore, if the target number of subjects has been enrolled, there is a possibility that additional subjects in screening may not be enrolled.

The study duration will include a 35-day maximum screening period; a 24-week randomized, double blind, parallel-group, active controlled treatment period, with 30-day and 70-day follow-ups if subjects are discontinued earlier or choose not to enter Period 2 (Period 1); and a 192-week open-label long term extension period with a 30-day follow-up call or site visit (Period 2).

Subjects who meet eligibility criteria will be randomized in a 1:1 ratio to one of two treatment groups:

- Group 1: Upadacitinib 15 mg QD, N = 275 (Period 1) → Upadacitinib 15 mg QD (Period 2)
- Group 2: Abatacept IV, N = 275 (Period 1) → Upadacitinib 15 mg QD (Period 2)

Randomization will be stratified by number of prior bDMARD use (stratum 1: failed 1 or 2 biologics of the same class; stratum 2: failed  $\geq$  3 biologics of the same class or failed biologics of multiple classes) AND geographic region.

Subjects must have been on stable csDMARD(s) treatment for  $\geq 4$  weeks prior to the first dose of study drug and must remain on a stable dose until Week 12; the csDMARD dose may be decreased only for safety reasons. Starting at Week 12 (after Week 12)



assessments have been performed), initiation of or change in corticosteroids, non-steroidal anti-inflammatory drugs (NSAIDs), acetaminophen, or adding or increasing doses for up to 2 csDMARDs (concomitant use of up to 2 csDMARDs except the combination of MTX and leflunomide) is allowed as per local label.

Rescue therapy will be offered to subjects who meet the following criteria:

• Starting at Week 12, subjects who do not achieve ≥ 20% improvement in both TJC and SJC at two consecutive visits will be rescued with optimizing (initiate or increase) background RA medications: NSAIDs, corticosteroids, low-potency analgesics, acetaminophen or adding or increasing doses in up to 2 csDMARDs (concomitant use of up to 2 csDMARDs except the combination of MTX and leflunomide) and, if necessary, a burst of systemic corticosteroids (prednisone equivalent ≤ 0.5 mg/kg/day for 3 consecutive days), intra-articular, intramuscular, intravenous, trigger point or tender point, intra-bursa, and intratendon sheath injections of corticosteroids, dosage and frequency per standard of care, are allowed.

Subjects who complete the Week 24 visit (end of Period 1) will enter the open-label long term extension portion of the study, Period 2 (192 weeks). Subjects who are assigned to upadacitinib 15 mg QD treatment group in Period 1 will continue to receive upadacitinib 15 mg QD per original randomization assignment. Subjects who are assigned to abatacept IV in Period 1 will be switched to receive upadacitinib 15 mg QD.

An unblinded analysis will be conducted after all subjects have completed Period 1 (Week 24). Period 2 is open-label.

Study design schematics of Period 1 and Period 2 are shown in Figure 1 and Figure 2, respectively.

Figure 1. Period 1 Study Design



csDMARD = conventional synthetic disease modifying anti-rheumatic drug; DMARD = disease modifying anti-rheumatic drug; n = number; QD = once daily; RA = rheumatoid arthritis; W = week

- \* The follow-up period is only for subjects who do not enter Period 2.
- \*\* Subjects randomized to Group 1 under Amendment 3 received 30 mg QD dose. Starting with Amendment 4, subjects randomized to Group 1 will receive 15 mg QD dose.

PERIOD 2:
Copen-Label Extension Period (192 Weeks)

Follow-Up Period (≈ 30 days)

Group 1:
Upadacitinib 15 MG
QD\*

Upadacitinib 15 MG
QD\*

Upadacitinib 15 MG
QD\*

Figure 2. Period 2 Study Design

QD = once daily; W = week

\* Subjects who enrolled under Amendment 3, including subjects on both upadacitinib and abatacept will continue to receive open-label upadacitinib 30 mg QD. Subjects who enroll under Amendment 4 or 3.01 or later will receive open-label upadacitinib 15 mg QD. Starting with Amendment 5, all subjects will receive open-label 15 mg QD, including those currently on upadacitinib 30 mg QD.

W32

W36

(and every 12 weeks)

W216

# 4.3 Study Design History

W24

W28

The study was originally designed to compare upadacitinib dose of 30 mg QD versus abatacept IV. In October 2017, the study protocol was amended (Amendment 4) to replace the upadacitinib 30 mg arm with the upadacitinib dose of 15 mg QD. This decision was made based on data from the initial, placebo controlled periods of the upadacitinib Phase 3 RA Studies M13-549 (csDMARD-IR) and M13-542 (bDMARD-IR). The data from these studies showed that both the 15 and 30 mg QD doses achieved superior responses to placebo for all primary and ranked secondary endpoints at Week 12



and 30 mg dose provided no incremental benefit over the 15 mg dose. Safety results from these studies showed that upadacitinib 15 mg and 30 mg QD doses were well-tolerated.

In Period 1, subjects randomized to upadacitinib arm under Amendment 3 received 30 mg QD dose. As such, 44 subjects in total were enrolled under Amendment 3. Starting with Amendment 4, new subjects randomized to upadacitinib arm will receive 15 mg QD dose. In Period 2, subjects who enrolled under Amendment 3, including subjects randomized to both Upadacitinib 30 mg QD and Abatacept IV, will receive open-label upadacitinib 30 mg QD; all subjects who enroll under Amendment 4 or thereafter will receive open-label upadacitinib 15 mg QD. Starting with Amendment 5, all subjects will receive open label upadacitinib 15 mg QD dose, including those currently on upadacitinib 30 mg QD.

The subjects enrolled before and after Protocol Amendment 4 form two separate cohorts and the cohort from Protocol Amendment 4 is considered the main cohort for the study. The statistical analyses for these two cohorts will be conducted differently as described in Section 5.1.

#### 4.4 Sample Size

The planned total sample size of 550 (N = 275 per arm) is applied to the cohort of upadacitinib 15mg QD vs abatacept IV that is enrolled after Protocol Amendment 4. This sample size can provide more than 90% power for the non-inferiority assessment on the primary endpoint using a non-inferiority margin of 0.6 at two-sided significance level of 0.05, assuming true difference between upadacitinib 15 mg QD and abatacept in change from baseline in DAS28 (CRP) at Week 12 is 0.5 with an assumed standard deviation of 2.0 and accounting for a 10% dropout rate. Under the planned sample size, superiority comparison of upadacitinib 15 mg QD to abatacept in change from baseline in DAS28 (CRP) is powered at approximately 80%. The planned sample size can also provide approximately 80% power for superiority comparison of upadacitinib 15 mg QD to abatacept in DAS28 (CRP) Clinical Remission (DAS28 (CRP) < 2.6) at two-sided significance level of 0.05 and accounting for a 10% dropout rate, where the assumed



DAS28 (CRP) CR response rate is 31% for upadacitinib 15 mg QD and for 20% abatacept.

## 4.5 Interim Analysis and Date Base Lock

An unblinded analysis will be conducted after all subjects have completed Period 1 (Week 24).

## 4.6 Data Monitoring Committee (DMC) Activities

An independent external Data Monitoring Committee (DMC) is used to review unblinded safety data at regular intervals during the conduct of the study as described in the DMC charter. The DMC will provide recommendation to an AbbVie Point of Contact on whether to continue, modify, or terminate studies after each review. When needed, high-level unblinded efficacy data may also be requested by the DMC and be reviewed so that the DMC can assess benefit:risk of any emerging safety differences.

# 5.0 Analysis Populations and Analysis Windows

# 5.1 Analysis Populations

The study contains two cohorts of subjects: the "30 mg Cohort" which includes the subjects randomized to Upadacitinib 30 mg QD vs Abatacept IV, and the "15 mg Cohort" which includes the subjects randomized to Upadacitinib 15 mg QD vs Abatacept IV. The 15 mg Cohort is the main cohort for statistical analysis. For the 30 mg Cohort, the full analysis set and safety analysis set are defined. For 15 mg Cohort, the full analysis set, per protocol analysis set and safety analysis set are defined.

For the 30 mg Cohort, no formal statistical analysis is planned. The scope of data reporting and the statistical methods for descriptive summary are provided in Appendix A.

The statistical analysis described in Chapters 6 to 10 applies to the 15 mg Cohort.



#### Full Analysis Set (FAS)

The Full Analysis Set (FAS) includes all randomized subjects who received at least one dose of study drug. The FAS will be used for all efficacy and baseline analyses.

#### Per Protocol Analysis Set

The Per Protocol Analysis Set represents a subset of the FAS and consists of all FAS subjects who did not meet any major protocol deviations that can potentially impact the Week 12 efficacy assessment. Additional analysis of the primary efficacy endpoint will be conducted on the Per Protocol analysis set, in order to evaluate the impact of major protocol deviations.

Major protocol deviations (ICH deviations and other clinically significant non-ICH deviations) will be identified prior to database lock.

# Safety Analysis Set

The Safety Analysis Set consists of all subjects who received at least one dose of study drug. For the Safety Analysis Set, subjects are assigned to a treatment group based on the "as treated" treatment group, regardless of the treatment randomized. The "as treated" is determined by the treatment the subject received during the majority of the subject's drug exposure time in the analysis period.

#### 5.2 Analysis Windows

#### **Definition of Study Days (Days Relative to the First Dose of Study Drug)**

Study Days are calculated for each collection date relative to the date of the first dose of study drug. It is defined as the number of days between the date of the first dose of study drug and the collection date. Study days are negative values when the collection date of interest is prior to the first study drug dose date. Study days are positive values when the collection date of interest is on or after the first study drug dose date. The day of the first dose of study drug is defined as Study Day 1, while the day prior to the first study drug



dose is defined as Study Day -1 (there is no Study Day 0). Study days are used to map actual study visits to the protocol-specified study visits.

#### **Definition of Analysis Windows**

The following rules will be applied to assign actual subject visits to protocol-specified visits. For each protocol-specified study visit, a target study day will be identified to represent the corresponding visit along with a window around the target day. Windows will be selected in a non-overlapping fashion so that a collection date does not fall into multiple visit windows. If a subject has two or more actual visits in one visit window, the visit closest to the target day will be used for analysis. If two visits are equidistant from the target day, then the later visit will be used for analysis.

The visit window and the target study day for each protocol-specified visit in Period 1 are displayed in Table 1, Table 2, Table 3, and Table 4 (depending on the different visit schedules of different endpoints). Visit windows for protocol-specified visits in Period 2 are defined similarly.

Table 1. Analysis Windows for Efficacy Analysis for Period 1 (for ACR Components and Morning Stiffness) and Safety Analysis for Period 1 (for Labs and Vital Signs)

| <b>Protocol Specified Visit Week</b> | <b>Lower Bound</b> | Target Day | <b>Upper Bound</b> |
|---|---|---|---|
| Baseline | -99 | 1ª | 1 |
| 2 | 2 | 15 | 22 |
| 4 | 23 | 29 | 43 |
| 8 | 44 | 57 | 71 |
| 12 | 72 | 85 | 99 |
| 16 | 100 | 113 | 127 |
| 20 | 128 | 141 | 155 |
| 24 | 156 | 169 | first dose date of Period 2 |

a. Day of first dose of study drug.

Table 2. Analysis Windows for Efficacy Analysis for Period 1 (for EQ 5D 5L and SF-36)

| <b>Protocol Specified Visit Week</b> | Lower Bound | Target Day | Upper Bound |
|---|---|---|---|
| Baseline | <b>-99</b> | 1ª | 1 |
| 4 | 2 | 29 | 57 |
| 12 | 58 | 85 | 127 |
| 24 | 128 | 169 | first dose date of Period 2 |

a. Day of first dose of study drug.

Table 3. Analysis Windows for Efficacy Analysis for Period 1 (for FACIT-F)

| <b>Protocol Specified Visit Week</b> | Lower Bound | Target Day | Upper Bound |
|---|---|---|---|
| Baseline | -99 | 1ª | 1 |
| 4 | 2 | 29 | 43 |
| 8 | 44 | 57 | 71 |
| 12 | 72 | 85 | 99 |
| 16 | 100 | 113 | 141 |
| 24 | 142 | 169 | first dose date of Period 2 |

a. Day of first dose of study drug.

Table 4. Analysis Windows for Efficacy Analysis for Period 1 (for WPAI)

| <b>Protocol Specified Visit Week</b> | Lower Bound | Target Day | Upper Bound |
|---|---|---|---|
| Baseline | -99 | 1ª | 1 |
| 4 | 2 | 29 | 43 |
| 8 | 44 | 57 | 71 |
| 12 | 72 | 85 | 127 |
| 24 | 128 | 169 | first dose date of Period 2 |

a. Day of first dose of study drug.

# 6.0 Demographics, Baseline Characteristics, Medical History, and Previous/Concomitant Medications

## 6.1 Demographics and Baseline Characteristics

Demographic and baseline characteristics information will be collected at the Baseline visit of the study and will be summarized for the FAS. The number of observations, mean, standard deviation, median, minimum and maximum will be summarized for continuous variables. Categorical or discrete variables will be summarized via frequencies and percentages. Summary statistics will be computed for each treatment group and overall.

#### Main Demographic and Baseline Characteristics

- Sex (male, female)
- Age (years)
- Age Categories ( $< 40, [40, 65], \ge 65 \text{ years}$ )
- Race (White, Black or African American, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, Asian, Other)
- Geographic Region (North America, South/Central America, Western Europe, Eastern Europe, Asia, Other)
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino)
- Weight (kg)
- Weight Categories ( $< 60 \text{ kg}, \ge 60 \text{ kg}$ )
- Height (cm)
- Body Mass Index (BMI) (kg/m2)
- Body Mass Index (BMI) Category (kg/m2) (BMI  $\leq$  25, BMI  $\geq$  25)

#### **RA Medical History and Characteristics**

- Duration of RA Symptoms in years
- Duration of RA Diagnosis in years



- Duration of RA Symptoms Categories ( $< 10 \text{ year}, \ge 10 \text{ year}$ )
- Duration of RA Diagnosis Categories ( $< 10 \text{ year}, \ge 10 \text{ year}$ )
- Number of prior bDMARD received  $(1, 2, \ge 3)$
- Prior failed bDMARD (stratum 1: failed 1 or 2 biologics with the same mechanism of action; stratum 2: failed ≥ 3 biologics with the same mechanism of action and/or multiple mechanisms of action)
- Failed at least one prior bDMARD due to lack of efficacy (yes, no)
- Failed at least one anti-TNF (yes, no)
- Oral steroid dose at baseline (yes, no)
- Oral steroid dose (prednisone equivalent) at baseline
- Concomitant csDMARD at baseline (MTX alone, MTX plus other csDMARD, csDMARD other than MTX)

#### ACR and/or DAS Components at Baseline

- Tender joint count (TJC68) defined as the number of tender joints out of 68 assessed joints
- Swollen joint count (SJC66) defined as the number of swollen joints out of 66 assessed joints
- Tender joint count (TJC28) defined as the number of tender joints out of 28 assessed joints used for DAS28 calculation
- Swollen joint count (SJC28) defined as the number of swollen joints out of 28 assessed joints used for DAS28 calculation
- Physician's global assessment of disease activity (mm on a 100-mm horizontal visual analogue scale [VAS])
- Patient's assessment of pain within last week (mm on a 100-mm horizontal VAS)
- Patient's global assessment of disease activity within last 24 hours (mm on a 100-mm horizontal VAS)
- Health Assessment Questionnaire Disability Index of the (HAQ DI) (range: 0 to 3)



- High sensitivity C-reactive protein (hsCRP) (mg/L)
- Erythrocyte sedimentation rate (ESR) (mm/hr)

#### Other Baseline RA Disease Characteristics

- Anti-cyclic citrullinated peptide (Anti-CCP) (units)
- Anti-CCP status: Positive or Negative
- Rheumatoid Factor (RF) (units)
- Rheumatoid Factor (RF) status: Positive or Negative
- RF and Anti-CCP both positive vs. at least one negative
- RF and Anti-CCP both negative vs. at least one positive
- DAS28 [hsCRP]
- DAS28 [ESR]
- DAS28 Categories:
  - o DAS28 > 5.1 (High Disease Activity)
  - $\circ$  DAS28  $\leq$  5.1
- Clinical Disease Activity Index (CDAI)
- CDAI categories:
  - CDAI > 22 (High Disease Activity)
  - o CDAI ≤ 22
- Simplified Disease Activity Index (SDAI)
- SDAI categories:
  - SDAI > 26 (High Disease Activity)
  - $\circ$  SDAI  $\leq 26$

### **Patient Report Outcomes at Baseline**

- Morning stiffness (severity and duration)
- EQ-5D-5L
- FACIT-F

- 36-Item Short Form Health Survey (SF-36) Version 2: physical component summary, mental component summary and the 8 sub-domain scores
- WPAI

#### **Clinical Tests at Screening**

- Chest x-ray
- ECG
- Tuberculin PPD skin test, QuantiFERON TB Gold test
- Hepatitis Testing
- Serum pregnancy test

## **Immunization History**

- BCG immunization
- Herpes Zoster immunization
- Hepatitis B immunization

#### **Tobacco/Nicotine and Alcohol Use**

- Tobacco/Nicotine Use [user, ex-user, non-user, unknown]
- Alcohol Use [drinker, ex-drinker, non-drinker, unknown]

## 6.2 Medical History

Medical history data will be summarized and presented for FAS population using body systems and conditions/diagnoses as captured on the CRF. The body systems will be presented in alphabetical order and the conditions/diagnoses will be presented in alphabetical order within each body system. The number and percentage of subjects with a particular condition/diagnosis will be summarized for each randomized treatment group as well as overall. Subjects reporting more than one condition/diagnosis within a body



system will be counted only once for that body system. No statistical comparison will be performed for medical history reporting.

#### 6.3 Prior Treatment and Concomitant Medications

Prior and concomitant medications will be summarized by each randomized treatment group as well as overall for FAS. Prior medications are those medications taken prior to the first dose of study drug. This includes medications with a start date before the first study drug administration date, regardless of the end date of these medications. Medications taken on the day of the first dose of study drug are not counted as prior medications. Concomitant medications are those medications, other than study drug, taken after the first dose of study drug and within 28 days of the last dose of study drug. This includes medications with a start date between first study drug administration and last study drug administration + 28 days, as well as, medications with a start date prior to first dose of study drug and which are ongoing after first dose of study drug. Medications taken on the day of the first dose of study drug are counted as concomitant medications.

The number and percentage of subjects who received a prior medication and the number and percentage of subjects who received a concomitant medication will be tabulated separately by the generic name assigned by the most current version of the World Health Organization (WHO) Drug Dictionary.

#### 6.4 Protocol Deviations

Protocol deviations based on ICH deviation criteria are categorized as follows:

- 1. Those who entered the study even though they did not satisfy the entry criteria
- 2. Those who developed withdrawal criteria during the study and were not withdrawn
- 3. Those who received the wrong treatment or incorrect dose, and
- 4. Those who received an excluded or prohibited concomitant medication.



The protocol deviations listed above will be summarized and listed by treatment group.

# 7.0 Patient Disposition

The following will be summarized by randomized treatment group as well as overall:

- number of subjects randomized,
- number of subjects included in key analysis populations (Full Analysis Set, Per Protocol Analysis Set for primary efficacy analysis, Safety Analysis Set for Period 1),
- number of subjects who completed Period 1 study participation,
- number of subjects who entered Period 2,
- number of subjects who completed overall study (Period 1 and Period 2) participation (if applicable).

This summary will be repeated by site.

Premature discontinuation details will be further summarized separately for Period 1 and Period 2 as follows.

### Period 1

The number and percentage of subjects completed Period 1 and prematurely discontinued in Period 1 will be summarized by randomized treatment group, separately by study drug and study participation completion/discontinuation, with the primary reason for discontinuation collected from CRF by the following categories:

- Adverse event (AE)
- Withdrew consent
- Lost to follow-up
- Lack of efficacy (this option is collected as a reason for study drug discontinuation, not for study participation discontinuation)
- Other



Subjects may have more than one reason for discontinuing, but only the primary reason will be summarized.

In addition, the number and percentage of subjects who entered Period 2 will also be summarized by randomized treatment group.

#### Period 2

Period 2 patient dispositions and reason for discontinuation will be summarized for the single treatment group Upadacitinib 15 mg QD in Period 2.

Among the subjects who entered Period 2 participation (regardless of whether subject is on study drug in Period 2), the number and percentage of subjects completed and prematurely discontinued study participation in Period 2 will be summarized. Among the subjects who entered Period 2 on study drug, the number and percentage of subjects completed and prematurely discontinued study drug in Period 2 will be summarized.

For subjects who prematurely discontinued study drug or study participation, the primary reason as well as all reasons for discontinuation will be summarized with the same categories as given above for Period 1.

# 8.0 Study Drug Exposure and Compliance

# 8.1 Study Drug Exposure

The duration of exposure to study drug will be summarized for the safety analysis set by the following groups.

- Upadacitinib 15 mg QD
   This includes Upadacitinib 15 mg QD exposure from subjects starting on
   Upadacitinib 15 mg QD and subjects switching from abatacept IV to Upadacitinib
   15 mg QD.
- 2. Abatacept IV

The duration of exposure to study drug will be summarized for each group as specified above, with the number of subjects, mean, standard deviation, median, minimum and maximum values. In addition, the number and percentage of subjects exposed to study drug will be summarized for the following cumulative duration intervals.

- $\geq 2$  weeks
- $\geq 1$  month
- $\geq$  3 months
- $\geq$  6 months
- $\geq 9$  months
- $\geq 12$  months
- $\bullet$  > 18 months
- $\geq 2$  years
- $\geq 2.5$  years
- $\geq 3$  years
- $\geq$  4 years

# 8.2 Compliance

Study drug compliance for upadacitinib 15 mg QD/PBO and for abatacept/PBO will be summarized separately for each treatment group for Period 1. Upadacitinib 15 mg QD/PBO compliance is defined as the number of upadacitinib 15 mg QD/PBO tablets taken (i.e., the difference between the number of tablets dispensed and the number of tablets returned) during Period 1 divided by the number of days that the subject was in the Treatment Phase in Period 1. Abatacept/PBO compliance is defined as the number of injections administered during the subject's participation in Period 1 divided by the number of injections planned during the subject's participation in the Treatment Phase in Period 1.

# 9.0 Efficacy Analysis

#### 9.1 General Considerations

There are two sets of planned efficacy analysis: efficacy analysis for Period 1 and long-term efficacy analysis. All efficacy analyses will be carried out using the FAS population.

# 9.1.1 Efficacy Analysis at Different Phases of the Study

#### **Efficacy Analysis for Period 1**

Standard efficacy analysis by randomized treatment groups (Upadacitinib 15 mg QD and Abatacept IV) will be performed on efficacy data for Period 1 (up to Week 24). No protocol-defined treatment switching will occur prior to the time point. Formal statistical inference will be generated, and results from this set of analysis will be used as the key efficacy findings of this study.

Long-Term Efficacy Analysis

Long-term efficacy analysis will be performed on As Observed data (defined in Section 9.1.2) by randomized treatment group sequence as described below:

- 1. Upadacitinib 15 mg QD
- 2. Abatacept IV → Upadacitinib 15 mg QD

There will be no statistical testing; only descriptive statistics and confidence intervals will be provided.

# 9.1.2 Definition of Missing Data Imputation

# Non-Responder Imputation (NRI) Approach

The NRI approach will categorize any subject who has a missing value for categorical variables at a specific visit as non-responder for that visit. In addition, subjects who



prematurely discontinue from study drug will be considered as non-responders for all subsequent visits after discontinuation.

### **Observed Cases (OC)**

The OC analysis will not impute values for missing evaluations. In addition, the OC will not use values after premature discontinuation of study drug. This sensitivity analysis will only be applied to the analysis in Period 1.

#### As Observed (AO)

The AO analysis will not impute values for missing evaluations. Regardless of treatment switching or premature discontinuation of study drug, all observed data will be used in the analysis. The AO analysis will be applied to long-term efficacy analysis.

#### **Multiple Imputation (MI)**

The MI analysis will impute missing data multiple times under appropriate random variation and thus generate multiple imputed "pseudo-complete" datasets. Results will be aggregated across the multiple imputed datasets, overcoming drawbacks of the single imputation methods. PROC MI will be used to generate 5 datasets using the fully conditional specification (FCS) method. Specifically, treatment group is included in the FCS imputation model to enable sampling stratified by treatment groups. Additionally, the imputation model includes demographics variables and baseline disease characteristics, as well as longitudinal response observed at any other visits. An ANCOVA model will first be performed on each of the multiple imputed datasets adjusting for treatment, stratification factor and baseline value. PROC MIANALYZE will then be used to aggregate the results for the final statistical inference using Rubin's method. The imputation is based on the assumption of data being missing at random. The missing at random assumption is considered reasonable given the high placebo response rate typically seen in RA trials. Additionally in RA trials, the proportion of discontinuation is relatively small (10-15% only) and the rate of discontinuation due to lack of efficacy is generally low (< 5%).



# <u>Mixed Effect Model Repeat Measurement (MMRM) and Generalized Linear Mixed Model (GLMM) for Long-Term Analysis</u>

The repeated measure analysis will be conducted using mixed model including As Observed measurements at all visits. MMRM will be used for continuous endpoints and GLMM will be used for binary endpoints. The mixed models will include the categorical fixed effects of treatment, visit and treatment-by-visit interaction, and main stratification factor prior bDMARD use. For the MMRM analysis of change from baseline in continuous endpoints, the baseline measurement will be included as a continuous fixed covariate. The categorical fixed effect of subject's discontinuation status may also be included in the model as appropriate. Unstructured, Toeplitz, compound symmetry, or other covariance structures may be considered.

# 9.2 Efficacy Analysis for Period 1

# 9.2.1 Primary Efficacy Analysis

The primary endpoint is the non-inferiority comparison of upadacitinib 15 mg QD to abatacept on change from baseline in DAS28 (CRP) at Week 12.

Analysis of the primary endpoint will be conducted on the FAS based on randomized treatment groups (Upadacitinib 15 mg QD and Abatacept IV). Statistical inference will be conducted using analysis of covariance (ANCOVA) coupled with MI for missing data handling. Specifically, the ANCOVA model will include treatment as the fixed factor, and the corresponding baseline value and the stratification factor of prior bDMARD use as the covariates. The LS mean and 95% CI will be reported for each randomized treatment group; the LS mean treatment difference and associated 95% CI will be reported comparing Upadacitinib 15 mg QD group and Abatacept IV group. The non-inferiority of Upadacitinib 15 mg QD versus Abatacept will be tested using the 95% confidence interval (CI) of treatment difference against a non-inferiority margin of 0.6.



### 9.2.2 Sensitivity Analysis of Primary Efficacy Variables

A sensitivity analysis will be conducted using ANCOVA based on Observed Cases without any imputation. This will be conducted on the FAS based on randomized treatment groups.

The primary analysis will be repeated on the Per Protocol Analysis Set as a supportive analysis.

# 9.2.3 Key Secondary Efficacy Analyses

Ranked key secondary endpoints (at Week 12) are:

- 1. Change from baseline in DAS28 (CRP) at Week 12 (superiority)
- 2. Proportion of subjects achieving DAS28 (CRP) Clinical Remission (CR) at Week 12 (superiority)

For the continuous endpoint change from baseline in DAS28 (CRP), the mean, standard deviation, median, and range will be reported for each randomized treatment group (Upadacitinib 15 mg QD and Abatacept IV). Statistical inference will be derived from the same analysis as the primary endpoint of the non-inferiority assessment using analysis of covariance (ANCOVA) coupled with MI for missing data handling, and p-value will be reported for the superiority comparison of Upadacitinib 15 mg QD versus Abatacept IV.

For the binary endpoint proportion of subjects achieving DAS28 (CRP) Clinical Remission (CR), frequencies and percentages will be reported for each randomized treatment group (Upadacitinib 15 mg QD and Abatacept IV). Point estimate and 95% CI using normal approximation will be provided for the response rate for each randomized treatment group. Point estimate, 95% CI and p-value will be provided for the treatment comparison between Upadacitinib 15 mg QD and Abatacept IV using the Cochran-Mantel-Haenszel test adjusting for the stratification factor of prior bDMARD use. NRI will be used as primary analysis and OC will be used as sensitivity analysis.



## 9.2.4 Exploratory Efficacy Analyses

Additional efficacy analysis includes the following endpoints at all visits in Period 1 unless specified otherwise:

- Proportion of subjects achieving DAS28 (CRP) LDA at Week 12 (non-inferiority with 10% margin);
- ACR20/50/70 response rates;
- Change from baseline in individual components of ACR response;
- Change from baseline in DAS28 (CRP) and DAS28 (erythrocyte sedimentation rate [ESR]);
- Change from baseline in SF-36 at Weeks 4, 12 and 24;
- Change from baseline in morning stiffness (severity and duration);
- Proportion of subjects achieving LDA or CR based on DAS28 (CRP), DAS28 (ESR), Simplified Disease Activity Index (SDAI), and Clinical Disease Activity Index (CDAI) criteria;
- Change from baseline in EQ-5D-5L at Weeks 4, 12 and 24;
- Change from baseline in Functional Assessment of Chronic Illness Therapy fatigue (FACIT-F) at Weeks 4, 8, 12, 16 and 24;
- Change from baseline in Work Productivity and Activity Impairment (WPAI) at Weeks 4, 8, 12 and 24;
- Change from baseline in CDAI and SDAI;
- Proportion of subjects achieving change from baseline in HAQ-DI  $\leq$  -0.3 and  $\leq$  -0.22, respectively;
- ACR/EULAR Boolean remission;
- Systemic corticosteroid dose from Week 12 to 24 (see Section 9.4.16 for details).

For binary endpoints, point estimate and 95% CI using normal approximation will be provided for the response rate for each randomized treatment group. Point estimate, 95% CI and p-value will be provided for the treatment comparison between Upadacitinib 15 mg QD and Abatacept IV using the Cochran-Mantel-Haenszel test adjusting for



stratification factor prior bDMARD use. The non-inferiority of Upadacitinib 15 mg QD versus Abatacept in DAS28 (CRP) LDA at Week 12 will be tested using the 95% confidence interval for treatment comparison against a non-inferiority margin of 10%. NRI will be used as primary analysis and OC will be used as sensitivity analysis.

For continuous endpoints, analysis will be conducted using ANCOVA based on Observed Cases without any imputation. The ANCOVA model will include treatment as the fixed factor, and the corresponding baseline value and the main stratification factors as the covariates. The LS mean and 95% CI will be reported for each randomized treatment group. The LS mean treatment difference and associated 95% CI and p-values between Upadacitinib 15 mg QD and Abatacept IV will be provided.

# 9.2.5 Handling of Multiplicity

In order to preserve the overall Type I error, a step-down approach will be used to test the primary and ranked key secondary endpoints where statistical significance can be claimed for a lower ranked endpoint only if the previous endpoint in the sequence meets the requirements of significance. Specifically, the testing will utilize the endpoint sequence of primary endpoint followed by ranked key secondary endpoints in the order as specified in Section 9.2.3, using two-sided  $\alpha$  of 0.05.

# 9.2.6 Efficacy Subgroup Analysis

The primary efficacy endpoint will be examined in the subgroups listed in Table 5 below. Treatment difference between Upadacitinib 15 mg QD and Abatacept IV will be presented with point estimate and 95% confidence interval using ANCOVA based on Observed Cases without imputation. No formal non-inferiority or superiority comparison will be performed at subgroup level. If any of the resulting subgroups has fewer than 10% of the planned study size (i.e., < 55 subjects), the subgroup analyses for that variable will not be presented.



**Table 5.** Insert Table Title Here

| Subgroup Factor | Categories |
|---|---|
| Age | < 40, 40 − < 65, ≥ 65 |
| Sex | Male or Female |
| Weight | $< 60 \text{ kg or} \ge 60 \text{ kg}$ |
| BMI | $< 25 \text{ or } \ge 25$ |
| Race | White, non-white |
| Geographic Region | North America, South/Central America, Western<br>Europe, Eastern Europe, Asia, Other |
| Duration of RA diagnosis | $< 10$ year or $\ge 10$ year |
| Baseline Rheumatoid Factor Status | Positive or Negative |
| Baseline Anti-CCP Antibody Status | Positive or Negative |
| Baseline both RF positive and Anti-CCP positive | Yes or No |
| Baseline both RF negative and Anti-CCP negative | Yes or No |
| Baseline DAS28 (CRP) | $\leq 5.1 \text{ or } > 5.1$ |
| Prior failed bDMARD | stratum 1: failed 1 or 2 biologics with the same mechanism of action; stratum 2: failed ≥ 3 biologics with the same mechanism of action and/or multiple mechanisms of action |
| Failed at least one Prior bDMARD due to lack of efficacy | Yes or No |
| Failed anti-IL6 due to lack of efficacy | Yes or No |

# 9.3 Long-Term Efficacy Analysis

Assessments to evaluate long-term efficacy will be analyzed for the following measures at each visit through Week 216 unless specified otherwise:

- ACR20/50/70 response rates;
- Change from baseline in individual ACR components;
- Change from baseline in DAS28 (CRP) and DAS28 (ESR);
- Change from baseline in SF-36 up to Week 48 only;
- Change from baseline in morning stiffness;

- Proportion of subjects achieving LDA based on DAS28 (CRP), DAS28 (ESR), SDAI, and CDAI criteria;
- Proportion of subjects achieving CR based on DAS28 (CRP), DAS28 (ESR), SDAI, and CDAI criteria;
- Change from baseline in EQ-5D-5L up to Week 48 only;
- Change from baseline in Functional Assessment of Chronic Illness Therapy fatigue (FACIT-F) up to Week 48 only;
- Change from baseline in Work Productivity and Activity Impairment (WPAI) at Week 48 only;
- Change from baseline in CDAI and SDAI;
- Proportion of subjects achieving a change from baseline in HAQ-DI  $\leq$  -0.3;
- Proportion of subjects achieving a change from baseline in HAQ-DI  $\leq$  -0.22;
- ACR/EULAR Boolean remission;
- Proportion of subjects with no concomitant corticosteroid use

Analyses will be based on As Observed (AO) data. Descriptive statistics will be provided for each randomized treatment group sequence as defined in Section 9.1.1. These include the number of observations, mean, standard deviation, and 95% CI for continuous endpoints; and frequencies and percentages with 95% CI using normal approximation for binary endpoints. In addition, longitudinal analysis will be performed using MMRM or GLMM as described in Section 9.1.2 for all endpoints except proportion of subjects with no concomitant corticosteroid use. Point estimates and 95% CI from the model will be provided for each treatment group sequence. Plot for each randomized treatment group sequence over time will be provided.

## 9.4 Efficacy Variables Definitions and Conventions

#### 9.4.1 ACR Criteria

ACR criteria are a commonly used standard criteria set mentioned in the guidance of American College of Rheumatology to evaluate the effectiveness of investigation drug in



RA clinical trials. It is a composite measurement calculated based on the improvement over a set of core measurements.

ACR20 is defined as at least 20% improvement (compared to baseline values) in tender and swollen joint counts and at least 20% improvement in 3 of the remaining 5 core set measures (subject global assessment of pain, subject global assessment of disease activity, physician global assessment of disease activity, subject assessment of physical function and acute phase reactant hsCRP).

ACR50 and ACR70 are similarly defined with at least 50% and 70% improvement, respectively.

A subject will be classified as an ACR20 (ACR50, ACR70) responder, if the following conditions are met:

- 1.  $\geq$  20% (50%, 70%) improvement from baseline in tender joint count (TJC68) and
- 2.  $\geq 20\%$  (50%, 70%) improvement from baseline in swollen joint count (SJC66) and
- 3.  $\geq 20\%$  (50%, 70%) improvement from baseline in at least 3 of the following 5:
  - patient's assessment of pain
  - patient's global assessment of disease activity (PGA)
  - physician's global assessment of disease activity (PhGA)
  - patient's self-assessment of physical function (i.e., measured by Health Assessment Questionnaire HAQ-DI score)
  - Acute-phase reactant value CRP

There are seven components to be evaluated to define an ACR response. Missing values for each component can occur due to a missed visit or due to dropout from the study. Depending on the pattern of the missing components, ACR responses may be or may not be determined using observed values only.

To maximize the utilization of observed information at certain visits and be scientifically as robust as possible, the principle to calculate ACR response is to minimize imputation whenever possible. Observed ACR response will be calculated first based on a derived visit window instead of the nominal visit identifier (e.g., Week 6 visit) collected from the CRF.

#### To calculate observed ACR responses:

- Identify the observed component xx% improvement indicator (0/1/missing), 1 means achieving  $\ge xx\%$  improvement from baseline and 0 means < xx% improvement from baseline (e.g., xx% representing 20%/50%/70%).
- ACRxx = 0 if TJC indicator = 0 OR SJC indicator = 0 OR at least 3 out of 5 components improvement indicators = 0.
- ACRxx = 1 if TJC indicator = 1 AND SJC indicator = 1 AND at least 3 out of 5 components improvement indicators = 1.
- For all other cases, ACRxx = missing since ACRxx cannot be determined.

The following table illustrates examples for ACR calculations.

| Example | TJC<br>68 | SJC<br>66 | Component 1 | Component 2 | Component 3 | Component 4 | Component 5 | ACR20-<br>Response? |
|---|---|---|---|---|---|---|---|---|
| A | 1 | 1 | 1 | 1 | 1 | | | Yes |
| В | 1 | 0 | 1 | 1 | 1 | 1 | 1 | No |
| C | | 0 | | | | | | No |
| D | 1 | | 1 | 1 | 1 | 1 | 1 | |
| E | 1 | 1 | 0 | 0 | 0 | 1 | 1 | No |
| F | | | 0 | 0 | 0 | | | No |
| G | 1 | 1 | 1 | 1 | 0 | 0 | • | |

Legend:  $1 = \ge 20\%$  improved compared to baseline; 0 = < 20% improved compared to baseline; "." = Missing

#### Windowing Rule for ACR Response Calculation:

• ACR component values will first be determined at each date within a visit window.



- ACR component values at each date will be combined to determine the observed ACR composite score at each date in each window.
- After this calculation, if multiple non-missing ACR composite scores are
  available within a given visit window, the non-missing ACR composite score
  closest to the target day will be used. If two composite scores have the same
  distance from the target day, the later one will be used. The corresponding date
  will be used as the observed ACR response date in the derived efficacy dataset.
- If a non-missing ACR composite score is not available for any day within a given visit window, the windowed component values for that visit will be used to calculate the ACR composite score for that visit window (component value windowing follow the same rules as in steps described above). The date of observed ACR composite score will be determined by the first available ACR component date, in the order of TJC, SJC, Pain, PGA, PhGA, HAQ-DI, CRP/ESR, in the derived efficacy dataset.

When observed ACR xx response for a given visit is missing, imputation methods will be used to calculate "imputed" ACRxx response.

- Non-Responder Imputation (NRI) for ACR response:
  - Step 1: all missing components will be imputed using LOCF, and then the ACR composite score can be calculated.
  - Step 2: if the ACR composite score cannot be determined by step 1, the ACR composite score will be imputed as 0. In addition, subjects who prematurely discontinue from the study drug will be considered as nonresponders (ACR = 0) for all subsequent visits after the discontinuation date.

#### 9.4.2 Joint Evaluation

Anatomical joints are evaluated for swelling and tenderness at every study visit. The 34 anatomical joints in Table 6 are assessed in this study for both the left and right side of the body.

Table 6. Anatomical Joints Assessed for Calculation of Tender and Swollen Joint Counts (TJC68 and SJC66)

| Temporomandibular | Sternoclavicular | Acromio-clavicular | Shoulder |
|---|---|---|---|
| Elbow | Wrist | Metacarpophalangeal I | Metacarpophalangeal II |
| Metacarpophalangeal III | Metacarpophalangeal IV | Metacarpophalangeal V | Thumb Interphalangeal |
| Proximal Interphalangeal<br>II | Proximal Interphalangeal<br>III | Proximal Interphalangeal IV | Proximal Interphalangeal<br>V |
| Distal<br>Interphalangeal II | Distal<br>Interphalangeal III | Distal<br>Interphalangeal IV | Distal<br>Interphalangeal V |
| Hip <sup>a</sup> | Knee | Ankle | Tarsus |
| Metatarsophalangeal I | Metatarsophalangeal II | Metatarsophalangeal III | Metatarsophalangeal IV |
| Metatarsophalangeal V | Great Toe/Hallux | Interphalangeal II | Interphalangeal III |
| Interphalangeal IV | Interphalangeal V | | |

a. Hip joints are not assessed for swelling.

At each study visit, a joint evaluator assessed whether a particular joint was "tender or painful" where presence of tenderness was scored as "1" and the absence of tenderness was scored as "0," provided the joint was not replaced ("9") or could not be assessed ("NA") due to other reasons (e.g., post-corticosteroid joint injection). The total tender joint count (TJC68), which is based on 68 joints, will be derived as the sum of all "1s" and proportional extrapolation will be used to impute joint counts for the joints that are replaced or not assessed. A similar method will be followed for the derivation of total swollen joint count (SJC66), which is based on 66 joints as the hip joints are excluded. Thus, the range for TJC68 will be 0 to 68 and 0 to 66 for SJC66.

# 9.4.3 Patient's Global Assessment of Disease Activity Visual Analog Scale (VAS)

The subject will assess his/her disease activity for the past 24 hours using a Patient's Global Assessment of Disease VAS. The range is 0 to 100 mm with no activity being indicated by 0 and severe activity by 100.
# 9.4.4 Physician's Global Assessment of Disease Activity Visual Analog Scale (VAS)

The physician will assess Patient's disease activity at the time of visit using a Physician's Global Assessment of Disease VAS. The range is 0 to 100 mm with no activity being indicated by 0 and severe activity by 100.

#### 9.4.5 Patient's Global Assessment of Pain

The subject will assess his/her pain in the previous week using a Patient's Global Assessment Pain VAS. The range is 0 to 100 mm with no pain being indicated by 0 and severe pain by 100.

### 9.4.6 Disease Activity Score (DAS28)

DAS28 (CRP) and DAS28 (ESR) are composite indices to assess disease activity in RA patients using hsCRP or ESR measurement respectively. The DAS provides a score between 0 and 10, indicating how active the rheumatoid arthritis is at the time of measurement.

DAS28 (CRP) and DAS28 (ESR) can be calculated based on Tender Joint Count, Swollen Joint Count, Patient's Global Assessment of Disease Activity (PtGA) (in mm), and hsCRP (in mg/L) or ESR (mm/hr).

DAS28 (CRP) = 
$$0.56 \times \sqrt{\text{(TJC28*)} + 0.28} \times \sqrt{\text{(SJC28**)} + 0.36} \times \ln(\text{hsCRP\&} + 1) + 0.014 \times \text{PtGA} + 0.96$$

DAS28 (ESR) = 
$$0.56 \times \sqrt{\text{(TJC28*)} + 0.28} \times \sqrt{\text{(SJC28**)} + 0.70} \times \ln(\text{ESR\#}) + 0.014 \times \text{PtGA}$$
»

- \* TJC28 refers to the Subject's total Tender Joint Count out of the provided 28 evaluated joints.
- \*\* SJC28 refers to the Subject's total Swollen Joint Count out of the provided 28 evaluated joints.
- & hsCRP refers to the high-sensitivity c-reactive protein lab value. hsCRP unit in the DAS28 (CRP) equation is expressed as mg/L.
- # ESR refers to the Erythrocyte sedimentation rate. ESR unit in the DAS28 (ESR) equation is expressed as mm/hr.
- » PtGA refers to the Patient's Global Assessment of Disease Activity.

where  $\sqrt{\ }$  is square root and  $\ln$  is natural  $\log$ .

Table 7. Anatomical Joints for DAS28 (CRP) Calculation

| Shoulder | Elbow | Wrist | Thumb Interphalangeal |
|---|---|---|---|
| Metacarpophalangeal I | Metacarpophalangeal II | Metacarpophalangeal III | Metacarpophalangeal IV |
| Metacarpophalangeal V | Proximal Interphalangeal<br>II | Proximal Interphalangeal<br>III | Proximal Interphalangeal IV |
| Proximal Interphalangeal<br>V | Knee | | |

To calculate observed DAS28 scores, the observed component value will be calculated first. Then the components will be included in the calculation per the DAS formula selected. If any observed component is missing in a window, then the observed DAS28 score will be missing.

### 9.4.7 Simplified Disease Activity Index (SDAI)

SDAI is a composite continuous index to assess disease activity based on TJC28, SJC28, Patient's Global Assessment of Disease Activity (PtGA) (in cm, 0 - 10), Physician's Global Assessment of Disease Activity (PhGA) (in cm, 0 - 10) and hsCRP (mg/dL). It can be derived as follows:

$$SDAI = TJC28 + SJC28 + PtGA (cm) + PhGA (cm) + hsCRP (mg/dL).$$

To calculate observed SDAI scores, the observed component value will be calculated first. Then the components will be included in the calculation per the SDAI formula selected. If any observed component is missing in a window, then the observed SDAI score will be missing.

### 9.4.8 Clinical Disease Activity Index (CDAI)

CDAI is a composite continuous index to assess disease activity without using hsCRP measurement. It can be calculated based on TJC28, SJC28, Patient's Global Assessment of Disease Activity (PtGA) (in cm, 0-10) and Physician's Global Assessment of Disease Activity (PhGA) (in cm, 0-10). It can be derived as follows:

CDAI = TJC28 + SJC28 + PtGA (cm) + PhGA (cm).

To calculate observed CDAI scores, the observed component value will be calculated first. Then the components will be included in the calculation per the CDAI formula selected. If any observed component is missing in a window, then the observed CDAI score will be missing.

### 9.4.9 Clinical Remission (CR) and Low Disease Activity (LDA)

Clinical remission (CR) and low disease activity (LDA) based on DAS28 (CRP), DAS28(ESR), SDAI and CDAI are defined as follows:

| | DAS28 (CRP) and DAS28 (ESR) | SDAI | CDAI |
|-----|-----------------------------|--------|-------|
| LDA | ≤ 3.2 | ≤ 11.0 | ≤ 10 |
| CR | < 2.6 | ≤ 3.3 | ≤ 2.8 |

#### 9.4.10 ACR/EULAR Boolean Remission

ACR/EULAR Boolean remission is defined based on the following four criteria:

- Tender joint count  $\leq 1$  (based on 28 joints)
- Swollen joint count  $\leq 1$  (based on 28 joints)
- $CRP \le 1 \text{ mg/dL}$
- Patient global assessment of disease activity  $\leq 10$  (mm)

All four criteria must be satisfied at a visit for a subject to be classified as achieving ACR/EULAR Boolean remission.

# 9.4.11 Disability Index of Health Assessment Questionnaire (HAQ DI)

HAQ-DI is a self-reported patient outcome measurement. It is calculated as the mean of the scores from 8 following categories with a range 0-3: Dressing and Grooming, Rising, Eating, Walking, Hygiene, Reach, Grip, and Activities. The higher the score, the more likely to associate with morbidity and mortality for the RA patient.

The maximum score for all the questions in each category is considered as the score for the category. The Standard disability index (HAQ-DI) takes into account the subject's use of aids or devices or assistance in the scoring algorithm for a disability category. For each of the eight disability categories there is an AIDS OR DEVICES companion variable(s) that is used to record the type of assistance, if any, a subject uses for his/her usual activities. If aids or devices and/or assistance from another person are checked for a disability category, the score for this category is set to 2 (much difficulty), if the original score is 0 (no difficulty) or 1 (some difficulty). The HAQ-DI is then calculated by summing the adjusted categories scores and dividing by the number of categories answered. The HAQ-DI cannot be calculated if the patient does not have scores for at least 6 categories.

### 9.4.12 EuroQoL-5D (EQ-5D-5L)

EQ-5D is a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D consists of 2 pages. The first page measures 5 dimensions of the health status (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) with 5 levels per dimension (no problems, slight problems, moderate problems, severe problems, and extreme problems corresponding to Level 1 to Level 5 respectively). The second page is an EQ Visual Analogue Scale (EQ VAS). EQ-5D health states, defined by the EQ-5D-5L descriptive system on the first page, may be converted into a single index value. The change from baseline of the index value and EQ VAS will be analyzed and reported. UK scoring algorithm will be used.

# 9.4.13 Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F)

Fatigue is one of the most frequent complaints of the elderly and is strongly associated with loss of independence and decreased physical activity and functional decline. One validated tool to measure fatigue is FACIT Fatigue Scale v4. The FACIT Fatigue Scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. Each of the fatigue and

impact of fatigue items are measured on a four point Likert scale. The FACIT Fatigue Scale is ranged from 0 to 52 and the higher the score, the better the quality of life. Score for each item is calculated by either subtracted from 4 or adding 0 depending on whether it is a reversal item or not. FACIT Fatigue Scale is then calculated by adding up all item scores, multiplied by 13 and divided by the number of items answered. It is essentially a prorated subscale if there are missing values for some items. If less than or equal to 50% of the items are answered (e.g., 6 out of 13), the proration is not acceptable and the scale will not be computed.

#### 9.4.14 Form SF-36v2

The 36-Item Short Form, Version 2 (SF-36v2) Questionnaire with 4 week recall will be completed by the subject at Baseline, Weeks 4, 8 and at study completion (Week 12 or at PD). The SF-36v2 health survey consists of 36 general health questions and this study is using the form for 4 weeks recall period (standard form). It has 2 components: physical and mental. For each component, a transformed summary score is calculated using 8 sub domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health.

The coding and scoring for the SF-36 will use the software provided by QualityMetrics.

### 9.4.15 Work Productivity and Activity Impairment (WPAI)

The Work Productivity and Activity Impairment (WPAI) questionnaire is a validated, self-administered tool used to assess the impact of disease on productivity. It measures time missed from work and impairment of work and activities due to a specific health problem. The questionnaire consists of 6 questions concerning a patient's ability to work and perform regular activities. Unemployed patients only answer select WPAI questions relating to their employment status and ability to perform daily activities other than work. WPAI scores are expressed as percent impairment based on six items. The four main impairment measures or scores are absenteeism, presenteeism, percent overall work impairment and percent activity impairment.



### 9.4.16 Systemic Corticosteroid Dose

This endpoint is to assess for differential corticosteroid use between treatment groups during the period between Week 12 and Week 24, due to Week 12 rescue criteria allowing dose changes with regard to corticosteroids. Systemic corticosteroid dose standardized by the duration of treatment phase, represented as average dose per day between Week 12 and Week 24, is calculated. The change from baseline dose to this average daily dose will be analyzed.

### 10.0 Safety Analysis

#### 10.1 General Considerations

Safety analyses will be carried out using the Safety Analysis Set. There are two sets of planned safety analysis: safety analysis for Period 1, and long-term safety analysis.

### **Safety Analysis For Period 1**

Standard safety analysis by the "as treated" treatment groups of Upadacitinib 15 mg QD and Abatacept IV will be performed on safety data up to Week 24. No protocol-defined treatment switching will occur prior to Week 24.

The standard safety analyses will include reporting of adverse events (AEs), laboratory, and vital signs measurements. Frequency tables of subjects with treatment-emergent adverse events (TEAEs) by system organ class (SOC) and by preferred term (PT) as in the Medical Dictionary for Regulatory Activities (MedDRA) dictionary will be provided by treatment group. Mean changes from baseline in all continuous laboratory parameters and vital signs variables at each visit will be summarized by "as treated" treatment group. Frequency tables of subjects meeting criteria for potentially clinically significant vital sign values and for potentially clinically significant laboratory values will be provided by treatment group. Missing safety data will not be imputed.



### **Long-Term Safety Analysis**

Long-term safety analyses for upadacitinib 15 mg QD include reporting of AE rate adjusted by cumulative exposure, mean change from baseline in laboratory parameters and vital sign variables, and rate of potentially clinically significant laboratory and vital signs values. The treatment-emergent adverse event (TEAE) rate per 100 patient-years of exposure will be presented. Listing of subjects with TEAEs by SOC and PT will be provided. Mean changes from baseline in all continuous laboratory parameters and vital signs variables at each visit will be summarized by "as treated" treatment group sequences defined as follows. Frequency tables and listings of subjects meeting criteria for potentially clinically significant vital sign values and for potentially clinically significant laboratory values will be provided. Missing safety data will not be imputed.

"As treated" treatment group sequences are defined as follows:

- 1. Upadacitinib 15 mg QD
- 2. Abatacept IV → Upadacitinib 15 mg QD

### 10.2 Analysis of Adverse Events

A treatment-emergent Adverse Event (TEAE) is defined as an adverse event with an onset date that is after the first dose of study drug, and no more than 30 days or 5 half-lives of the drug, whichever is larger, after the last dose of study drug. Specifically, 30 days will be used for Upadacitinib 15mg QD, and 70 days will be used for abatacept.

Events where the onset date is the same as the study drug start date are assumed to be treatment-emergent, unless the study drug start time and the adverse event start time are collected and the adverse event start time is prior to the study drug start time. If an incomplete onset date was collected for an adverse event, the event will be assumed to be treatment-emergent unless there is other evidence that confirms that the event was not treatment-emergent (e.g., the event end date was prior to the study drug start date).



Adverse event data will be presented by SOCs and PTs using MedDRA Version 21.0 or most up to date version, in which adverse events will be sorted in alphabetical order by SOC and PT.

### 10.2.1 Analysis of Adverse Events for Period 1

### 10.2.1.1 Adverse Events Overview

The number and percentage of subjects experiencing TEAEs will be summarized by "as treated" treatment group for the following AE categories.

- All TEAEs
- Treatment-emergent serious adverse events (SAEs)
- Treatment-emergent severe adverse events
- TEAEs reasonably possibly related to study drug
- TEAEs of special interest
- TEAEs leading to discontinuation of study drug
- TEAE leading to death

In the AE overview summary, any event with an unknown severity will be considered as severe and any AE with an unknown relationship will be considered as having "reasonable possibility" of being related to study drug.

Additional AEs may be considered for tabulation/summary based on recommendations from Clinical and Safety as deemed appropriate.

For TEAEs of special interest, the point estimate and 95% CI (using normal approximation) will be provided for the treatment difference in AE percentage.

As a sensitivity analysis, the AE overview summary and AE of special interest overview summary will be repeated in which all AEs with an onset date after the first dose of study drug will be included, regardless of whether the AE occurred more than 30 days (or 70 days) after the last dose of study drug.



### 10.2.1.2 Adverse Events by System Organ Class and Preferred Term

The number and percentage of subjects experiencing adverse events will be tabulated by SOC and MedDRA PT by "as treated" treatment group. The SOCs will be presented in alphabetical order, and the PTs will be presented in alphabetical order within each SOC.

The following summaries of adverse events will be generated:

- All TEAEs
- Treatment-emergent serious adverse events (SAEs)
- Treatment-emergent severe adverse events
- TEAEs reasonably possibly related to study drug
- TEAEs leading to discontinuation of study drug
- TEAE leading to death
- Frequent AEs (reported in 2% of subjects or more in any treatment group)

Subjects reporting more than one adverse event for a given MedDRA preferred term will be counted only once for that term (most severe incident for the severity tables and most related incident for the relationship tables). Subjects reporting more than one type of adverse event within a SOC will be counted only once for that SOC. Subjects reporting more than one type of adverse event will be counted only once in the overall total.

As a sensitivity analysis, the AE summary by SOC and PT will be repeated, in which all AEs with an onset date after the first dose of study drug will be included, regardless of whether the AE occurred more than 30 days (or 70 days) after the last dose of study drug.

### 10.2.1.3 TEAEs by Maximum Severity

TEAEs will also be summarized by maximum severity by "as treated" treatment group. If a subject has an AE with an unknown severity, then the subject will be counted in the severity category of unknown, even if the subject has another occurrence of the same event with a severity present. The only exception is that if the subject has another



occurrence of the same AE with the most extreme severity – severe. In this case, the subject will be counted under the severe category.

### 10.2.1.4 TEAEs by Relationship

TEAEs will also be summarized by relationship to study drug, as assessed by the investigator, by "as treated" treatment group. If a subject has a TEAE with an unknown relationship, then the subject will be counted in the relationship category of "unknown," even if the subject has another occurrence of the same event with a relationship present. The only exception is if the subject has another occurrence of the same TEAE with a relationship assessment of "reasonable possibility." In this case, the subject will be counted under the "reasonable possibility" category.

# 10.2.1.5 Frequent (≥ 2%) Adverse Events and Reasonably Possibly Related Adverse Events by System Organ Class and Preferred Term

TEAEs and reasonably possibly related AEs occurring for more than 2% of the subjects in any of the "as treated" treatment groups will be summarized by MedDRA PT in decreasing frequency separately.

### 10.2.1.6 Adverse Events of Special Interest

The Adverse Events of Special Interest (AESI) categories will be summarized and presented by "as treated" treatment group using SOC and MedDRA PT. The AESI categories will be identified by the following search criteria per Standard MedDRA Queries (SMQs)/Company MedDRA Queries (CMQs) in Table 8 below. Adjudicated cardiovascular events will be summarized and presented by treatment group using the CAC adjudicated categories.



Table 8. AESI for Upadacitinib with SMQs/CMQs/PTs Searches

| AESI | Type of<br>MedDRA<br>Query | Broad or<br>Narrow<br>Search | SMQ/CMQ Search Criteria |
|---|---|---|---|
| Serious Infections | CMQ | | "Infections" – Subset for SAEs |
| Opportunistic Infection<br>excluding Tuberculosis and<br>Herpes Zoster | CMQ | | "Opportunistic Infection excluding<br>Tuberculosis and Herpes Zoster" |
| Possible Malignancy | SMQ | Narrow | "Malignancies" |
| Malignancy | SMQ | | "Malignant tumours" |
| Non-Melanoma Skin Cancer (NMSC) | SMQ | Narrow | Skin Malignant tumours (Narrow SMQ) removing Melanoma CMQ |
| Malignancy excluding NMSC | | | "Malignant tumours" SMQ removing NMSC output |
| Lymphoma | SMQ | | "Malignant Lymphomas" |
| Hepatic Disorder | SMQ | Narrow | "Drug Related Hepatic Disorders" |
| Adjudicated Gastrointestinal<br>Perforations | Output from adjudication | | |
| Anemia | CMQ | | "Non-Hemolytic and Non-Aplastic<br>Anemias" |
| Neutropenia | CMQ | | "Hematological Toxicity - Neutropenia" |
| Lymphopenia | CMQ | | "Hematological Toxicity - Lymphopenia" |
| Herpes Zoster | CMQ | | "Herpes Zoster" |
| Creatine Phosphokinase (CPK)<br>Elevation | PT | | Search only for the PT of "Blood creatine phosphokinase increased" |
| Renal Dysfunction | SMQ | Narrow | "Acute Renal, Failure" |
| Active Tuberculosis | CMQ | | "Active Tuberculosis" |
| Adjudicated Cardiovascular<br>Events | Output from CAC | | |
| MACE* | | | |
| Cardiovascular Death | | | |
| Non-fatal Myocardial<br>Infarction | | | |
| Non-fatal Stroke | | | |



**Table 8.** AESI for Upadacitinib with SMQs/CMQs/PTs Searches (Continued)

| AESI | Type of<br>MedDRA<br>Query | Broad or<br>Narrow<br>Search | SMQ/CMQ Search Criteria |
|---|---|---|---|
| Undetermined/Unknown<br>Cause of Deaths | | | |
| Other Cardiovascular events | | | |
| Adjudicated Thrombotic Events | Output From CAC | | |
| Venous Thromboembolic<br>Events** | | | |
| Deep Vein Thrombosis | | | |
| Pulmonary Embolism | | | |
| Other Venous Thrombosis | | | |
| Arterial Thromboembolic<br>Events (non-cardiac, non-<br>neurologic) | | | |

 $CAC = Cardiovascular\ Adjudication\ Committee;\ CMQ = company\ MedDRA\ query;\ PT = preferred\ term; \\ SMQ = standard\ MedDRA\ query$ 

- \* MACE; Major Adverse Cardiovascular Events, defined as cardiovascular death, non-fatal myocardial infarction and non-fatal stroke.
- \*\* Venous thromboembolic events (VTE) include deep vein thrombosis (DVT) and pulmonary embolism (PE) (fatal and non-fatal).

Additional AEs may be considered for tabulation/summary based on recommendations from Clinical and Safety as deemed appropriate.

### 10.2.2 Analysis of Long-Term Adverse Event Rates

Long-term adverse event rates for upadacitinib 15 mg QD will be analyzed using event rates adjusted by cumulative exposure. This includes TEAEs occurred under Upadacitinib 15 mg QD exposure from subjects starting on Upadacitinib 15 mg QD and subjects switching from Abatacept IV to Upadacitinib 15 mg QD.

For this event rate calculation, 1 year will be considered to be 365.25 days. For each treatment group, the numerator of the overall rate will be the total number of TEAEs



reported for the event; that is, a subject can contribute more than one event to the numerator. The denominator of the rates will be the total number of days exposed to upadacitinib 15 mg QD summed across all treated subjects divided by 365.25. The TEAE rate per 100 patient-years of exposure will be calculated as ([numerator/denominator])\*100. The number of TEAEs reported (numerator), the total number of years of study drug exposure (denominator), and the TEAE rate per 100 patient-years will be presented.

# 10.2.2.1 Overview of Adverse Events Rates per 100 Patient-Years of Study Drug Exposure

An overview of AEs per 100 patient-years of study exposure will be presented for the following AE categories.

- All TEAEs
- Treatment-emergent serious adverse events (SAEs)
- Treatment-emergent severe adverse events
- TEAEs reasonably possibly related to study drug
- TEAEs of special interest
- TEAEs leading to discontinuation of study drug
- TEAE leading to death

In the AE overview summary, any event with an unknown severity will be considered as severe and any AE with an unknown relationship will be considered as having "reasonable possibility" of being related to study drug.

Additional AEs may be considered for tabulation/summary based on recommendations from Clinical and Safety as deemed appropriate.



# 10.2.2.2 Adverse Events Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT

The TEAE rate per 100 patient-years of exposure will be calculated overall, for each SOC and each PT, for each of the following events:

- All TEAEs
- Treatment-emergent serious adverse events (SAEs)
- Treatment-emergent severe adverse events
- TEAEs reasonably possibly related to study drug
- TEAEs leading to discontinuation of study drug
- TEAE leading to death

# 10.2.2.3 Adverse Events of Special Interest Rates per 100 Patient Years of Study Drug Exposure

The Adverse Events of Special Interest (AESI) rate per 100 patient-years of exposure as outlined in Section 10.2.2 will be calculated overall, for each SOC and each PT, for each of the AESI listed in Section 10.2.1.6. Adjudicated cardiovascular events will be summarized and presented using the CAC adjudicated categories.

# 10.2.2.4 Listing of Serious Adverse Events (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation

All serious adverse events (SAEs), deaths, and adverse events leading to discontinuation of study drug will be listed.

### 10.3 Analysis of Laboratory Data

#### 10.3.1 Variables and Units

All laboratory parameters to be collected in this study are listed below. Laboratory parameters will be reported using the standard international (SI) units.



## Table 9. List of Laboratory Variables

Bicarbonate

| Laboratory Variables |
|---|
| Hematology |
| White Blood Cell (WBC) Count |
| Red Blood Cell (RBC) Count |
| Hemoglobin |
| Hematocrit |
| Platelets count |
| Neutrophils |
| Basophils |
| Eosinophils |
| Lymphocytes |
| Monocytes |
| Bands |
| Chemistry |
| Total Bilirubin |
| Alkaline Phosphatase (ALP) |
| Serum glutamic oxaloacetic transaminase/aspartate aminotransferase (SGOT/AST) |
| Serum glutamic pyruvic transaminase/alanine aminotransferase (SGPT/ALT) |
| Total Protein |
| Albumin |
| Glucose |
| Triglycerides |
| Blood Urea Nitrogen (BUN) |
| Creatinine |
| Uric acid |
| Sodium |
| Potassium |
| Calcium |
| Inorganic Phosphorus |
| Creatine Phosphokinase (CPK) |
| Chloride |

### **Table 9.** List of Laboratory Variables (Continued)

| Laboratory Variables |
|-------------------------------------|
| Chemistry (Continued) |
| Cholesterol (TC) |
| LDL cholesterol (LDL-C) |
| HDL cholesterol (HDL-C) |
| LDL-C/HDL-C ratio |
| TC/HDL-C ratio |
| Urinalysis |
| Specific Gravity |
| pH |
| Protein |
| Glucose |
| Ketones |
| Blood |
| Microscopic Examination (if needed) |
| Urobilinogen |
| Bilirubin |
| Leukocytes |
| Nitrites |
| Other |
| hs-CRP |
| QuantiFERON-TB Golda |
| IgG and IgM |
| DOD |

a. For annual follow-up QFT is captured only for those with negative QFT at Screening.

**ESR** 

# 10.3.2 Analysis of Laboratory Data for Period 1

The laboratory data will be summarized by the "as treated" treatment groups (Upadacitinib 15 mg QD and Abatacept IV).



# 10.3.2.1 Assessment of Mean Change from Baseline and Percentage Change from Baseline in Clinical Laboratory Variables

Analyses of mean change from baseline in continuous hematology, chemistry, and urinalysis variables which are measured longitudinally will be performed by visits and by "as treated" treatment group. For each change from baseline analysis, the following summary statistics will be presented for each treatment group: sample size, baseline mean, visit mean, and the mean, standard deviation, and median of the changes from baseline.

In addition, similar analyses will be conducted for percentage change from baseline in LDL-C, HDL-C, total cholesterol, triglycerides, and hemoglobin.

# 10.3.2.2 Assessment of Shift from Baseline in Clinical Laboratory Variables

The baseline and post-baseline laboratory observations will be categorized as Grade 1, Grade 2, Grade 3, and Grade 4 according to OMERACT criteria (Rheumatology Common Toxicity Criteria v.2.0). For creatine phosphokinase and creatinine, NCI CTC criteria will be used.

For each laboratory variable, shift tables will be generated that cross tabulate the subjects' as deemed appropriate by "as treated" treatment group:

- Category of the baseline value versus category of the final value.
- Category of the baseline value versus maximum category.
- Category of the baseline value versus minimum category.

Note that the minimum/maximum category is used, rather than the category of the minimum/maximum value. The two may be different due to variation in the reference range.

No statistical tests will be performed for this analysis.



# 10.3.2.3 Assessment of Potentially Clinical Significant Laboratory Values

The criteria for potentially clinically significant laboratory values will be determined by OMERACT criteria of Grade 3 or 4. For creatine phosphokinase and creatinine, NCI CTC criteria will be used.

The number and percentage of subjects meeting the criteria for potentially clinically significant laboratory values will be summarized by "as treated" treatment group. Only subjects with worsening in grade compared to baseline grade will be captured.

#### 10.3.2.4 Assessment of Liver Elevations

According to FDA's Guidance for Industry "Drug-Induced Liver Injury: Premarketing clinical evaluation" (July 2009), when aminotransferase (AT) abnormalities indicating hepatocellular injury are accompanied by evidence of impaired hepatic function (bilirubin elevation > 2 × ULN), in the absence of evidence of biliary obstruction (i.e., significant elevation of ALP) or some other explanation of the injury (e.g., viral hepatitis, alcohol hepatitis), the combined finding (i.e., Hy's Law cases) represents a signal of a potential for the drug to cause severe DILI.

For the purpose of assessing for potential Hy's law cases, the frequencies and percentages of subjects with post baseline liver specific function test values that meet the following criteria of potential clinical interest will be summarized by "as treated" treatment group:

- ALT  $> 3 \times ULN$
- ALT  $\geq$  5 × ULN
- ALT > 10 × ULN
- ALT  $\geq 20 \times ULN$
- AST  $\geq 3 \times ULN$
- $AST > 5 \times ULN$
- AST  $\geq 10 \times ULN$
- AST  $\geq 20 \times ULN$



- $TBL > 2 \times ULN$
- Alkaline phosphatase  $\geq 1.5 \times ULN$
- ALT and/or AST  $\geq$  3 × ULN and concurrent TBL  $\geq$  1.5 × ULN
- ALT and/or AST  $\geq 3 \times ULN$  and concurrent TBL  $\geq 2 \times ULN$

### 10.3.3 Analysis of Long-Term Laboratory Data

# 10.3.3.1 Assessment of Mean Change from Baseline and Percentage Change from Baseline in Clinical Laboratory Variables

Analyses of mean change from baseline in continuous hematology, chemistry, and urinalysis variables which are measured longitudinally will be performed by visits and by "as treated" treatment group sequences as described in Section 10.1. For each change from baseline analysis, the following summary statistics will be presented for each treatment group sequence: sample size, baseline mean, visit mean, and the mean, standard deviation, and median of the changes from baseline.

In addition, similar analyses will be performed for percentage change from baseline in LDL-C, HDL-C, triglycerides and hemoglobin.

# 10.3.3.2 Assessment of Potentially Clinically Significant Laboratory Values

Long-term laboratory data will be summarized based on the number and percentage of subjects meeting the criteria for potentially clinically significant laboratory values for upadacitinib 15 mg QD.

In the evaluation of potentially clinically significant laboratory values, the baseline value will be determined by the last non-missing measurement recorded on or before the date of the first dose of upadacitinib 15mg QD (which may be different than the first dose of study drug in the study). For example, for a subject who started on abatacept and switched to upadacitinib 15 mg QD, lab values under upadacitinib 15 mg QD exposure



would be evaluated against the baseline value defined as the last non-missing measurement recorded on or before the date of the first dose of upadacitinib 15 mg QD.

A listing of all subjects with any laboratory determination meeting OMERACT criteria of Grade 3 or 4 will be provided. For creatine phosphokinase and creatinine, NCI CTC criteria will be used. Only subjects with worsening in grade compare to baseline grade will be captured. For each of these subjects, the whole course of the respective parameter will be listed.

#### 10.3.3.3 Assessment of Liver Elevations

The frequencies and percentages of subjects with post-baseline liver-specific function test values that meet the criteria of potential clinical interest (as described in Section 10.3.2.4) will be summarized for upadacitinib 15 mg QD, similarly as described in Section 10.2.2.

A listing of potentially clinically significant liver elevations based on criteria specified above will be provided. For each of these subjects, the whole course of the respective parameter will be listed.

### 10.4 Analysis of Vital Signs

### 10.4.1 Variables and Criteria Defining Abnormality

Vital sign variables include sitting systolic blood pressure, sitting diastolic blood pressure, pulse rate, respiratory rate, body temperature, and weight. The criteria for potentially clinically significant vital sign findings are presented in Table 10.

Table 10. Criteria for Potentially Clinically Significant Vital Sign Findings

| Vital Sign | Category | Criteria for Potential Clinically Significant Vital Signs |
|---|---|---|
| Systolic blood pressure | Low | Value ≤ 90 mmHg and decrease ≥ 20 mmHg from Baseline |
| | High | Value $\geq 160$ mmHg and increase $\geq 20$ mmHg from Baseline |
| Diastolic blood pressure | Low | Value ≤ 50 mmHg and decrease ≥ 15 mmHg from Baseline |
| | High | Value $\geq 105$ mmHg and increase $\geq 15$ mmHg from Baseline |
| Weight | High | > 7% increase from baseline |
| | Low | > 7% decrease from baseline |

### 10.4.2 Analysis of Vital Sign for Period 1

Analyses of mean change from baseline in continuous vital sign variables which are measured longitudinally will be performed by visits and by the "as treated" treatment groups of Upadacitinib 15 mg QD and Abatacept IV. For each change from baseline analysis, the following summary statistics will be presented for each treatment group: sample size, baseline mean, visit mean, and the mean, standard deviation, and median of the changes from baseline.

The number and percentage of subjects meeting the criteria for potentially clinically significant vital sign values will be summarized by "as treated" treatment group.

### 10.4.3 Analysis of Long-Term Vital Sign

Analyses of mean change from baseline in continuous vital signs variables which are measured longitudinally will be performed by visits and by "as treated" treatment group sequences as described in Section 10.1. For each change from baseline analysis, the following summary statistics will be presented for each treatment group sequence: sample size, baseline mean, visit mean, and the mean, standard deviation, and median of the changes from baseline.

Long-Term Vital Sign will also be summarized based on the number and percentage of subjects meeting the criteria for potentially clinical significant vital sign for upadacitinib 15 mg QD. In the evaluation of potentially clinically significant vital sign values, the



baseline value will be determined by the last non-missing measurement recorded on or before the date of the first dose of upadacitinib 15 mg QD, similarly as described in Section 10.3.3.2.

A listing of all subjects with any vital sign values meeting the criteria for potentially clinically significant vital signs will be provided. For each of these subjects, the whole course of the respective parameter will be listed.

### 11.0 Summary of Changes

# 11.1 Summary of Changes between the Previous Version and the Current Version

The primary efficacy analysis and Period 1 reporting have been completed under the SAP version 1.0. The current SAP update applies only to future reporting of long-term analysis.

- 1. Updated to align with Protocol Amendment 5 and 6, including handling of dose switch from upadacitinib 30 mg QD to 15 mg QD for the 30 mg Cohort (Appendix A) and change of study length from 260 to 216 weeks.
- 2. Updated Section 9.1.2 to describe the missing data handling approach for the additional sensitivity analysis using longitudinal models for long-term efficacy.
- 3. Updated Section 9.3 to incorporate the additional sensitivity analysis for long-term efficacy.
- 4. Added language to clarify analysis details in Section 10.2.1.1, and Section 10.2.2.1.
- 5. Updated Section 10.2.1.6 and Section 10.4.1 to align with the latest upadacitinib AESI definitions in PSSAP V4.0.
- 6. Added Appendix B to describe analysis accounting for impact of COVID-19 pandemic.
- 7. Added Section 11.0 for summary of changes and Section 12.0 for SAP version history summary.

# 12.0 Version History

### **Table 11. SAP Version History Summary**

| Version | Date | Summary |
|---|---|---|
| 1.0 | 04 Jun 2019 | Original version. Version 1.0 was used for the primary analysis. |
| 2.0 | 17 Dec 2020 | Updated to align with Protocol Amendment 5 and 6, including handling of dose switch from upadacitinib 30 mg QD to 15 mg QD for the 30 mg Cohort and change of study length from 5 years to 216 weeks. Included additional sensitivity analysis for long-term efficacy, and analyses due to COVID-19 impact. |

# 13.0 Appendix

Appendix A Statistical Analysis for 30 mg Cohort

Appendix B Statistical Analysis to Account for Impact of COVID-19 Pandemic

Appendix C OMERACT Criteria



### **Appendix A.** Statistical Analysis for the 30 mg Cohort

For subjects in the 30 mg Cohort, descriptive summaries will be provided as follows.

### **Patient Disposition**

For subject accountability, by-site summary will be provided for each randomized treatment group (i.e., Upadacitinib 30 mg QD and Abatacept IV) for all the items described in the first paragraph of Section 7.0. Premature discontinuation details will be further summarized separately for Period 1 and Period 2, similar to as described in Section 7.0.

### Summary of Dose Switch from Upadacitinib 30 mg QD to 15 mg QD

Starting with Amendment 5, all subjects will receive open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 mg QD. The visit at which dose switch occurs could be different for each subject. For subjects in the 30 mg Cohort, the number and percentage of subjects switching to upadacitinib 15 mg QD at each visit will be summarized.

#### **Efficacy Analysis**

Descriptive summaries will be provided for DAS28 (CRP) change from baseline and Clinical Remission (CR) based on DAS28 (CRP) by randomized treatment group for Period 1 or by randomized treatment sequence for long term analysis as described below. Other efficacy data will be reported as collected in CSR 16.2 listings.

- Randomized treatment group sequence for long term analysis for the 30 mg
   Cohort: Abatacept IV → Upadacitinib 30 mg QD
- 2. Upadacitinib 30 mg QD

Starting with Amendment 5, all subjects will receive open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 mg QD. For long-term efficacy analysis,



subjects will continue to be summarized under the treatment sequences as described above, regardless of dose switch – i.e., data collected after dose switch will continue to be summarized under the same treatment sequences. The visit at which dose switch occurs could be different for each subject. The first and last visits at which dose switch occurs will be noted in the summary.

#### **Safety Analysis**

Safety analysis for the 30 mg Cohort includes Period 1 safety analysis and long-term safety analysis.

Period 1 safety analysis by the "as treated" treatment groups of Upadacitinib 30 mg QD and Abatacept IV will be performed up to Week 24. Period 1 safety analyses include the overview of treatment emergent adverse events (TEAE), overview of treatment emergent AESI and the TEAE summary by SOC and PT (similar to as described in Section 10.2.1.1 and Section 10.2.1.2).

For long-term safety analysis, adverse event rates for upadacitinib 30 mg QD will be summarized using event rates adjusted by cumulative exposure. Starting with Amendment 5, all subjects will receive open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 mg QD. For subjects who previously received upadacitinib 30 mg QD, adverse events and exposure to upadacitinib 30 mg QD will be censored at the time of dose switch; subsequent adverse events and exposure starting the day of first dose of upadacitinib 15 mg QD will be summarized under a separate group:

### 1. Upadacitinib 30 mg QD

This includes AEs occurred under Upadacitinib 30 mg QD exposure from subjects starting on Upadacitinib 30 mg QD and subjects switching from Abatacept IV to Upadacitinib 30 mg QD. Exposure is censored at time of dose switch from Upadacitinib 30 mg QD to Upadacitinib 15 mg QD.

2. Upadacitinib 15 mg QD switched from any Upadacitinib 30mg QD



This includes Upadacitinib 15 mg QD exposure from subjects who switched dose from Upadacitinib 30 mg QD to Upadacitinib 15 mg QD

Long term safety analysis will only include overview of TEAE rates per 100 patient-years of study drug exposure, overview of treatment emergent AESI event rates per 100 patient-years of study drug exposure, and the TEAE rate per 100 patient-years summary by SOC and PT (similar to as described in Section 10.2.2.1 and Section 10.2.2.2).

Additional long-term safety analysis for the any abatacept group, including abatacept subjects in both 15 mg Cohort and 30 mg Cohort, will be conducted. Specifically, overview of TEAE rates per 100 patient-years of study drug exposure, overview of treatment emergent AESI event rates per 100 patient-years of study drug exposure, and the TEAE rate per 100 patient-years summary by SOC and PT will be conducted.



### Appendix B. Statistical Analysis to Account for Impact of COVID-19 Pandemic

#### 1.0 Overview

The COVID-19 pandemic is interfering with the conduct of many ongoing trials, with potential impacts on treatment duration and collection, analysis and the interpretation of clinical trial data. Some protocol-specified visits in the clinical trials may be impacted due to COVID-19 infection or logistical restrictions during the pandemic. For example, some scheduled visits may be missed due to self-quarantine or local government restrictions on travel; some visits may also be delayed or canceled due to healthcare resource constraints during the pandemic. Impacted visits due to COVID-19 will be recorded in the database.

This appendix describes the additional analyses and updates to existing analyses due to COVID-19 impact. At the time of COVID-19 pandemic, all study subjects are in Period 2 of the study. The primary efficacy analysis and Period 1 reporting have been completed in 2019 and are not affected by the COVID-19 pandemic. The analyses described in this appendix are only applicable to Period 2 and future reporting of the long-term analyses.

### 2.0 Patient Disposition

Period 2 patient disposition and reason for discontinuation will be summarized as described in Section 7.0. For subjects who prematurely discontinued study drug or study participation, the reasons for discontinuation will be summarized with two additional categories capturing discontinuation due to COVID-19 infection or logistical restrictions related to the COVID-19 pandemic (as collected in CRF):

- Adverse event (AE)
- Withdrew consent
- Lost to follow-up
- Lack of efficacy
- COVID-19 infection
- COVID-19 logistical restrictions



#### • Other

In addition, the number and percentage of subjects with scheduled study visits affected by COVID-19 pandemic will be summarized by treatment group sequences. The impact on study visits will be summarized by the following categories (as collected in CRF) by visit:

- Missed visit
- Virtual visit
- In person, partial assessments done

### 3.0 Long Term Efficacy Analysis

Missing data could occur due to various reasons, including missing visits/assessments, early withdrawal from the study, or missing due to COVID-19 infection or logistic restriction. The probability of having missed visits and missing data due to COVID-19 infection or logistical restrictions related to the COVID-19 pandemic can be reasonably assumed to be unrelated to the unobserved values. Therefore, for the purpose of statistical analysis, it is reasonable to assume that these missing data are missing at random (MAR) and the statistical models that require MAR assumption are appropriate.

As described in Section 9.1.2, longitudinal analysis models MMRM and GLMM will be used for long term efficacy analysis and will be maintained for long term efficacy analysis in the presence of missing data due to COVID-19.

### 4.0 Safety Analysis

In listings of adverse events and deaths, a flag indicating whether the event or death was related to COVID-19 infection will be presented. A listing of COVID-19 related adverse events may be provided.



### Appendix C. OMERACT Criteria

| Rheumatology | Common | Toxicity | Criteria | v.2.0 |
|--------------|--------|----------|----------|-------|

Based on Woodworth TG, et al. Standardizing assessment of adverse effects in rheumatology clinical trials II. Status of OMERACT Drug Safety Working Group May 2006: OMERACT 8. Standardizing Assessment and Reporting of Adverse Effects in Rheumatology Clinical Trials: Enabling Description of Comparative Safety Profiles for Antirheumatic Therapies

| Safety Profiles for Antirheumatic Therapies | | | | |
|---|---|---|---|---|
| | 1 – Mild | 2 – Moderate | 3 – Severe | 4 – Includes Life Threatening |
| | Asymptomatic, or transient | Symptomatic | Prolonged symptoms, reversible, | At risk of death |
| | Short duration (< 1 week) | Duration (1 – 2 weeks) | major functional impairment | Substantial disability, especially if |
| | No change in life style | Alter lifestyle occasionally | Prescription meds/partial relief | permanent. |
| | No medication or OTC | Meds relieve. (may be | May be hospitalized < 24 hr | Multiple meds |
| | | prescription), | Temporary study drug | Hospitalised > 24 hr |
| | | Study drug continued | discontinuation, or/and dose reduced | Study drug discontinued |
| A. Allergic/Immunolo | ogic | | | |
| A1. Allergic reaction/ hypersensitivity (includes drug fever) | Transient rash: drug fever < 38°C: transient, asymptomatic bronchospasm | Generalised urticaria responsive to meds; or drug fever > 38°C, or reversible bronchospasm | Symptomatic bronchospasm requiring meds; symptomatic urticaria persisting with meds, allergy related oedema/angioedema | Anaphylaxis, laryngeal/pharyngeal oedema, requiring resuscitation |
| A2. Autoimmune reaction | Seriologic or other evidence of<br>autoimmune reaction, but patient<br>asymptomatic: all organ function<br>normal and no treatment is<br>required (e.g., vitiligo) | Evidence of autoimmune reaction involving a non-essential organ or functions, requiring treatment other than immunosuppressive drugs (e.g., hypothyroidism) | Reversible autoimmune reaction involving function of a major organ or toxicity requiring short term immunosuppressive treatment (e.g., transient colitis or anaemia) | Causes major organ dysfunction, or<br>progressive, not reversible, or<br>requires long-term administration<br>of high dose immunosuppressive<br>therapy |
| A3. Rhinitis<br>(includes sneezing,<br>nasal stuffiness, post-<br>nasal discharge) | Transient, non-prescription meds relieve | Prescription med. required, slow | Corticosteroids or other prescription med. with persistent disabling symptoms such as impaired exercise tolerance | NA |

| A4. Serum sickness | Transient, non-prescription meds relieve | Symptomatic, slow response to meds (e.g., oral corticosteroids) | Prolonged; symptoms only partially relieved by meds; parenteral corticosteroids required | Major organ dysfunction, requires long-term high-dose immunosuppressive therapy |
|---|---|---|---|---|
| A5. Vasculitis | Localised, not requiring treatment; or rapid response to meds; cutaneous | Symptomatic, slow response to meds (e.g., oral corticosteroids) | Generalised, parenteral corticosteroids required or/and short duration hospitalisation | Prolonged, hospitalisation, ischemic changes, amputation |
| B. Cardiac | | | | |
| B1. Arrhythmia | Transient, asymptomatic | Transient, but symptomatic or recurrent, responds to meds | Recurrent/persistent; maintenance prescription | Unstable, hospitalisation required, parenteral meds |
| B2. Cardiac function decreased | Asymptomatic decline in resting ejection fraction by > 10%, but < 20% of baseline value | Asymptomatic decline of resting ejection fraction ≥ 20% of baseline value | CHF responsive to treatment | Severe or refractory CHF |
| B3. Edema | Asymptomatic (e.g., 1 + feet/calves), self-limited, no therapy required | Symptomatic (e.g., 2 + feet/calves), requires therapy | Symptoms limiting function (e.g., 3 + feet/calves, 2 + thighs), partial relief with treatment prolonged | Anasarca; no response to treatment |
| B4. Hypertension<br>(new onset or<br>worsening) | Asymptomatic, transient increase<br>by > 20 mmHg (diastolic) or to<br>> 150/100 if previously normal,<br>no therapy required | Recurrent or persistent increase > 150/100 or by > 10 mmHg (diastolic), requiring and responding readily to treatment | Symptomatic increase > 150/100,<br>> 20 mmHg, persistent, requiring<br>multi agency therapy, difficult to<br>control | Hypertensive crisis |
| B5. Hypotension<br>(without underlying<br>diagnosis) | Transient, intermittent,<br>asymptomatic, orthostatic<br>decrease in blood pressure<br>> 20 mmHg | Symptomatic, without interference with function, recurrent or persistent > 20 mmHg decrease, responds to treatment | Syncope or symptomatic, interferes with function, requiring therapy and sustained medical attention, dose adjustment or drug discontinuation | Shock |
| B6. Myocardial ischaemia | Transient chest pain/ECG changes; rapid relief with nitro | Recurring chest pain, transient<br>ECG ST-T changes; treatment<br>relieves | Angina with infarction, no or minimal functional compromise, reduce dose or discontinue study drug | Acute myocardial infarction, arrthymia or/and CHF |

| B7. Pericarditis/<br>pericardial effusion | Rub heard, asymptomatic | Detectable effusion by<br>echocardiogram, symptomatic<br>NSAID required | Detectable on chest x-ray,<br>dyspnoea; or pericardiocentesis;<br>requires corticosteroids | Pulsus alternates with low cardiac output; requires surgery |
|---|---|---|---|---|
| B8. Phlebitis/thrombosis/ Embolism (excludes injection sites) | Asymptomatic, superficial, transient, local, or no treatment required | Symptomatic, recurrent, deep vein thrombosis, no anticoagulant therapy required | Deep vein thrombosis requiring anticoagulant therapy | Pulmonary embolism |
| C. General (constitut | ional) | | , | |
| C1. Fatigue/malaise (asthenia) | Increase over baseline; most usual daily functions maintained, short term | Limits daily function intermittently over time | Interferes with basic ADL, persistent | Unable to care for self, bed or wheelchair bound > 50% of day debilitating, hospitalisation |
| C2. Fever (pyrexia)<br>(note: fever due to<br>drug allergy should<br>be coded as allergy) | Transient, few symptoms 37.7 – 38.5°C | Symptomatic, recurrent 38.6 – 39.9°C. Relieved by meds | ≥ 40°C; ≤ 24 h, persistent symptoms; partial response to meds | ≥ 40°C, debilitating, > 24 h, hospitalisation; no relief with meds |
| C3. Headache | Transient or intermittent, no meds or relieved with OTC | Persistent, recurring, non-narcotic analgesics relieve | Prolonged with limited response to narcotic medicine | Intractable, debilitating, requires parenteral meds |
| C4. Insomnia | Difficulty sleeping, short term, no interfering with function | Difficulty sleeping interfering with function, use of prescription med | Prolonged symptoms, with limited response to narcotic meds | Debilitating, hospitalisation; no relief with meds |
| C5. Rigors, chills | Asymptomatic, transient, no meds, or non-narcotic meds relieve | Symptomatic, narcotic meds relieve | Prolonged symptoms, with limited response to narcotic meds | Debilitating, hospitalisation; no relief with meds |
| C6. Sweating (diaphoresis) | Episodic, transient | Frequent, short term | Frequent, drenching, disabling | Dehydration, requiring IV fluids/hospitalization > 24 hrs |
| C7. Weight gain | 5% – 9.9% | 10% – 19.9% | 20% – 30% | NA |
| C8. Weight loss | 5% – 9.9% | 10% – 19.9% | 20% - 30% | NA |

| D. Dermatologic | | | | |
|---|---|---|---|---|
| D1. Alopecia | Subjective, transient | Objective, fully reversible | Patchy, wig used, partly reversible | Complete, or irreversible even if patchy |
| D2. Bullous eruption | Localised, asymptomatic | Localised, symptomatic, requiring treatment | Generalised, responsive to treatment; reversible | Prolonged, generalised, or requiring hospitalisation for treatment |
| D3. Dry skin | Asymptomatic, controlled with emollients | Symptoms eventually (1 – 2 wks) controlled with emollients | Generalised, interfering with ADL > 2 wks, persistent pruritis, partially responsive to treatment | Disabling for extended period,<br>unresponsive to ancillary therapy<br>and requiring study drug<br>discontinuation for relief |
| D4. Injection site reaction | Local erythema, pain, pruritis, < few days | Erythema, pain, oedema, may include superficial phlebitis, 1 – 2 wks | Prolonged induration, superficial ulceration; includes thrombosis | Major ulceration necrosis requiring surgery |
| D5. Petechiae (without vasculitis) | Few, transient asymptomatic | Dependent areas, persistent up to 2 wks | Generalised, responsive to treatment; reversible | Prolonged, irreversible, disabling |
| D6. Photosensitivity | Transient erythema | Painful erythema and oedema requiring topical treatment | Blistering or desquamation, requires systematic corticosteroids | Generalised exfoliation or hospitalisation |
| D7. Pruritis | Localised, asymptomatic, transient, local treatment | Intense, or generalised, relieved by systematic medication | Intense or generalised; poorly controlled despite treatment | Disabling, irreversible |
| D8. Rash (not bullous) | Erythema, scattered<br>macular/popular eruption; pruritis<br>transient; TOC or no meds | Diffuse macular/popular eruption or erythema with pruritus; dry desquamation; treatment required | Generalised, moist desquamation, requires systemic corticosteroids; responsive to treatment; reversible | Exfoliative or ulcerating; or requires hospitalisation; or parenteral corticosteroids |
| D9.<br>Induration/fibrosis/<br>Thickening (not<br>sclerodermal) | Localized, high density on<br>palpation, reversible, no effect on<br>ADL and not disfiguring | Local areas < 50% body surface,<br>not disfiguring, transient<br>interference with ADL, reversible | Generalized, disfiguring, interferes with ADL, reversible | Disabling, irreversible, systemic symptoms |
| E. Ear/Nose/Throat | | | | |
| E1. Hearing loss | Transient, intermittent, no interference with function | Symptomatic, treatment required, reversible | Interferes with function; incomplete response to treatment | Irreversible deafness |

| E2. Sense of smell | Slightly altered | Markedly altered | Complete loss, reversible | Complete loss, without recovery |
|---|---|---|---|---|
| E3. Stomatitis | Asymptomatic | Painful, multiple, can eat | Interferes with nutrition, slowly reversible | Requires enteral support; residual dysfunction |
| E4. Taste<br>disturbance<br>(dysgeusia) | Transiently altered; metallic | Persistently altered; limited effect on eating | Disabling, effect on nutrition | NA |
| E5. Tinnitus | Intermittent, transient, no interference with function | Requires treatment, reversible | Disabling, or associated with hearing loss | Irreversible deafness |
| E6. Voice changes<br>(includes hoarseness,<br>loss of voice,<br>laryngitis) | Intermittent hoarseness, able to vocalise | Persistent hoarseness, able to vocalise | Whispered speech, slow return of ability to vocalise | Unable to vocalize for extended |
| E7. Xerostomia (dry mouth) | Transient dryness | Relief with meds | Interferes with nutrition, slowly reversible | Extended duration interference with nutrition, requires parenteral nutrition |
| F. Eye/Ophthalmolog | gic | | | |
| F1. Cataract | Asymptomatic, no change in vision, non-progressive | Symptomatic, partial visual loss, progressive | Symptoms impairing function, vision loss requiring treatment, including surgery | NA |
| F2. Conjunctivitis | Asymptomatic, transient, rapid response to treatment | Symptomatic, responds to treatment, changes not interfering with function | Symptoms prolonged, partial response to treatment, interferes with function | NA |
| F3. Lacrimation increased (tearing, watery eyes) | Symptoms not requiring treatment, transient | Symptomatic, treatment required, reversible | Unresponsive to treatment with major effect on function | NA |
| F4. Retinopathy | Asymptomatic, non-progressive, no treatment | Reversible change in vision; readily responsive to treatment | Disabling change in vision ophthalmological findings reversible, sight improves over time | Loss of sight |

| F5. Vision changes<br>(e.g., blurred,<br>photophobia, night<br>blindness, vitreous<br>floaters) | Asymptomatic, transient, no treatment required | Symptomatic, vision changes not interfering with function, reversible | Symptomatic, vision changes interfering with function | Loss of sight |
|---|---|---|---|---|
| F6. Xerophtalmia (dry eyes) | Mild scratchiness | Symptomatic without interfering with function, requires artificial tears | Interferes with vision/function, corneal ulceration | Loss of sight |
| G. Gastrointestinal | | | | |
| G1. Anorexia | Adequate food intake, minimal weight loss | Symptoms requiring oral nutritional supplementation | Prolonged, requiring iv support | Requires hospitalization for nutritional support |
| G2. Constipation | Asymptomatic, transient, responds to stool softener, OTC laxatives | Symptomatic, requiring prescription laxatives, reversible | Obstipation requiring medical intervention | Bowel obstruction. Surgery required |
| G3. Diarrhea | Transient, increase of 2 – 3 stools/day over pre-treatment (no blood or mucus), OTC agents relieve | Symptomatic, increase 4 – 6 stools/day, nocturnal stools, cramping, requires treatment with prescription meds | Increase > 6 stools/day, associated with disabling symptoms, e.g., incontinence, severe cramping, partial response to treatment | Prolonged, dehydration,<br>unresponsive to treatment, requires<br>hospitalization |
| G4. Dyspepsia (heartburn) | Transient, intermittent, responds to OTC antacids, H-2 blockers | Prolonged, recurrent, requires prescription meds, relieved by meds | Persistent despite treatment,<br>interferes with function, associated<br>with GI bleeding | NA |
| G5. GI bleed<br>(gastritis, gastric or<br>duodenal ulcer<br>diagnosed-define<br>aetiology) | Asymptomatic, endoscopic finding, haemocult + stools, no transfusion, responds rapidly to treatment | Symptomatic, transfusion ≤ 2 units needed; responds to treatment | Haematemesis, transfusion 3 – 4 units, prolonged interference with function | Recurrent, transfusion > 4 units, perforation, requiring surgery, hospitalisation |
| G6. Haematochezia (rectal bleeding) | Haemorrhodial, asymptomatic, no transfusion | Symptomatic, transfusion ≤ 2 units, reversible | Recurrent, transfusion > 3 – 4 units | > 4 units, hypotension, requiring hospitalization |

| G7. Hepatitis | Laboratory abnormalities, asymptomatic, reversible | Symptomatic laboratory<br>abnormalities, not interfering with<br>function, slowly reversible | Laboratory abnormalities persistent > 2 wks, symptoms interfere with function | Progressive, hepato-renal, anasarca, pre-coma or coma |
|---|---|---|---|---|
| G8. Nausea, or nausea/vomiting (use diagnostic term) | Transient, intermittent, minimal interference with intake, rapid response to meds | Persistent, recurrent, requires prescription meds, intake maintained | Prolonged, interferes with daily function and nutritional intake, periodic iv fluids | Hypotensive, hospitalization, parenteral nutrition, unresponsive to out-patient management |
| G9. Pancreatitis | Anylase elevation, intermittent nausea/vomiting, transient, responds rapidly to treatment | Amylase elevation with abdominal pain, nausea, occasional vomiting, responsive to treatment | Severe, persistent abdominal pain<br>with pancreatitic enzyme elevation,<br>incomplete or slow response to<br>treatment | Complicated by shock,<br>haemorrhage (acute circulatory<br>failure) |
| G10. Proctitis | Perianal pruritus, haemorrhoids<br>(new onset), transient, or<br>intermittent, relieved by OTC<br>meds | Tenesmus or ulcerations, anal fissure, responsive to treatment, minimal interference with function | Unresponsive to treatment, marked interference with function | Mucosal necrosis with<br>haemorrhage, infection, surgery<br>required |
| H. Musculoskeletal | | | | |
| H1. Avascular necrosis | Asymptomatic MRI changes, non-progressive | MRI changes and symptoms responsive to rest and analgesia | MRI changes, symptoms requiring surgical intervention | Wheelchair bound; surgical repair not possible |
| H2. Arthralgia | Intermittent transient symptoms, no meds or relieved by OTC meds | Persistent or recurrent symptoms, resolve with meds, little effect on function | Severe symptoms despite meds impairs function | Debilitating, hospitalisation required for treatment |
| H3. Leg cramps | Transient, intermittent, does not interfere with function | Recurrent symptoms, minimally interferes with function or sleep, responds to meds | Persistent, prolonged interference<br>with function or sleep, partial or no<br>response to meds | NA |
| H4. Myalgia | Occasional; does not interfere with function | Frequent, requires meds (non-<br>narcotic); minor effects on<br>function | Major change in function/lifestyle, narcotic pain meds | Debilitating, profound weakness, requires wheelchair, unresponsive to meds |

| I. Neuropsychiatric | | | | |
|---|---|---|---|---|
| I1. Anxiety or<br>Depression (mood<br>alteration) | Symptomatic, does not interfere with function; no meds | Frequent symptoms, responds to meds; interferes with ADL at times | Persistent, prolonged symptoms, partial or no response to meds, limits daily function | Suicidal ideation or danger to self |
| I2. Cerebrovascular ischaemia | NA | Single transient ischaemic event, responsive to treatment | Recurrent transient ischaemic events | Cerebrovascular vascular accident with permanent disability |
| I3. Cognitive disturbance | Subjective symptoms, transient, intermittent, not interfering with function | Objective symptoms, persisting, interferes with daily function occasionally | Persistent, or worsening objective symptoms; interferes with routine daily routine | Debilitating/disabling and permanent; toxic psychosis |
| I4. Depressed consciousness (somnolence) | Observed, transient, intermittent, not interfering with function | Somnolence or sedation, interfering with function | Persistent, progressive, obundation, stupor | Coma |
| I5. Inability to concentrate | Subjective symptoms, does not interfere with function | Objective findings, interferes with function | Persistent, prolonged objective findings or organic cause | NA |
| I6. Insomnia (in absence of pain) | Occasional difficulty sleeping,<br>transient intermittent, not<br>interfering with function | Recurrent difficulty sleeping;<br>requires meds for relief; occasional<br>interference with function | Persistent or worsening difficulty sleeping; severely interferes with routine daily function | NA |
| I7. Libido decreased | Decrease in interest | Loss of interest; influences relationship | Persistent, prolonged interfering with relationship | NA |
| I8. Peripheral motor<br>neuropathy | Subjective or transient loss of deep tendon reflexes; function maintained | Objective weakness, persistent, no significant impairment of daily function | Objective weakness with substantial impairment of function | Paralysis |
| I9. Peripheral sensory neuropathy (sensory disturbance) | Subjective symptoms without objective findings, transient, not interfering with function | Objective sensory loss, persistent, not interfering with function | Prolonged sensory loss or paraethesias interfering with function | NA |
| I10. Seizure | NA | Recurrence of old seizures, controlled with adjustment of medication | Recurrence/exacerbation with partial response to medication | Recurrence not controlled, requiring hospitalization; new seizures |

| I11. Vertigo (dizziness) | Subjective symptoms, transient, intermittent, no treatment | Objective findings, recurrent, meds relieve, occasionally interfering with function | Persistent, prolonged, interfering with daily function; partial response to medication | Debilitating without response to medication, hospitalization |
|---|---|---|---|---|
| J. Pulmonary | | | | |
| J1. Asthma | Occasional wheeze, no interference with activities | Wheezing, requires oral meds, occasional interference with function | Debilitating, requires nasal O <sub>2</sub> | Requires ventilator assistance |
| J2. Cough | Transient, intermittent, occasional OTC meds relieve | Persistent, requires narcotic or other prescription meds for relief | Recurrent, persistent coughing spasms without consistent relief by meds, interferes with function | Interferes with oxygenation; debilitating |
| J3. Dyspnea | Subjective, transient, no interference with function | Symptomatic, intermittent or recurring, interferes with exertional activities | Symptomatic during daily routine activities, interferes with function, treatment with intermittent nasal O <sub>2</sub> relieves | Symptomatic at rest, debilitating, requires constant nasal O <sub>2</sub> |
| J4. Pleuritic pain<br>(pleurisy) | Transient, intermittent symptoms, no treatment or OTC meds relieve | Persistent symptoms, requires prescription meds for relief | Prolonged symptoms, interferes with function, requires frequent narcotic pain relief | Debilitation, requiring hospitalisation |
| J5. Pneumonitis<br>(pulmonary<br>infiltrates) | Asymptomatic radiographic changes, transient, no treatment required | Symptomatic, persistent, requiring corticosteroids | Symptomatic, requiring treatment including O <sub>2</sub> | Debilitating, not reversible; or requiring assisted ventilation |
| J6. Pulmonary<br>function decreased<br>(FVC or carbon<br>monoxide diffusion<br>capacity – DLCO) | 76% – 90% of pre-treatment value | 51% – 75% of pre-treatment value | 26% – 50% of pre-treatment value | ≤ 25% of pre-treatment value |

| Laboratory Data | | | | |
|---|---|---|---|---|
| K. Haematology | | | | |
| K1. Hgb (g/dl)<br>decrease from pre-<br>treatment | 1.0 – 1.4 | 1.5 – 2.0 | 2.1 - 2.9, or Hgb $< 8.0$ , $> 7.0$ | ≥ 3.0; or Hgb < 7.0 |
| K2. Leukopenia<br>(total WBC) × 1000 | 3.0 – 3.9 | 2.0 – 2.9 | 1.0 – 1.9 | < 1.0 |
| K3. Neutropenia (× 1000) | 1.5 – 1.9 | 1.0 – 1.4 | 0.5 – 0.9 | < 0.5 |
| K4. Lymphopenia (× 1000) | 1.5 – 1.9 | 1.0 – 1.4 | 0.5 – 0.9 | < 0.5 |
| K5. Platelets (× 1000) | 75 – LLN | 50 – 74.9 | 20 – 49.9; platelet transfusion required | < 20; recurrent platelet transfusions |
| L. Chemistry | | | | |
| L1. Hypercalcaemia (mg/dl) | 1.1 × ULN – 11.5 | 11.6 – 12.5 | 12.6 – 13.5; or symptoms present | > 13.5; or associated coma |
| L2. Hyperglycemia (mg/dl) Fasting | 140 – 160 | 161 – 250 | 251 – 500 | > 500, or associated with ketoacidosis |
| L3. Hyperkalaemia (mmol/l)*** | 5.5 – 5.9 | 6.0 – 6.4 | 6.5 – 7.0 or any ECG change | > 7.0 or any arrhythmia |
| L5. Hypocalcaemia (mg/dl) | 0.9 × LLN – 7.8 | 7.7 – 7.0 | 6.9 – 6.5; or associated with symptoms | < 6.5 or occurrence of tetany |
| L6. Hypoglycemia (mg/dl) | 55 – 64 (no symptoms) | 40 – 54 (or symptoms present) | 30 – 39 (symptoms impair function) | < 30 or coma |
| L7. Hyponatraemia (mmol/l)*** | - | 125 – 129 | 120 – 124 | < 120 |

| L8. Hypokalaemia (mg/dl)*** | - | 3.0 – 3.4 | 2.5 – 2.9 | < 2.5 |
|---|---|---|---|---|
| L9. CPK (also if polymyositis-disease) | 1.2 – 1.9 × ULN | 2.0 – 4.0 × ULN | 4.0 × ULN with weakness but<br>without life-threatening signs or<br>symptoms | > 4.0 × ULN with signs or<br>symptoms of rhabdomyolysis or<br>life-threatening |
| L10. Serum uric acid | 1.2 – 1.6 × ULN | $1.7 - 2.9 \times ULN$ | $3.0 - 5.0 \times ULN$ or gout | NA |
| L11. Creatinine (mg/dl) | 1.1 – 1.3 × ULN | 1.4* – 1.8 × ULN | $1.9 - 3.0 \times ULN$ | > 3.0 × ULN |
| L12. SGOT (AST) | 1.2 – 1.5 × ULN | 1.6 – 3.0 × ULN | $3.1 - 8.0 \times ULN$ | > 8.0 × ULN |
| L13. SGPT (ALT) | 1.2 – 1.5 × ULN | 1.6 – 3.0 × ULN | $3.0 - 8.0 \times ULN$ | > 8.0 × ULN |
| L14. Alkaline phosphatase | 1.1 – 1.5** × ULN | 1.6 – 3.0 × ULN | $3.0 - 5.0 \times ULN$ | > 5.0 × ULN |
| L15. T. bilirubin | 1.1 – 1.4 × ULN | 1.5 – 1.9 × ULN | $2.0 - 3.0 \times ULN$ | > 3.0 × ULN |
| L16. LDH | $1.3 - 2.4 \times ULN$ | 2.5 – 5.0 × ULN | 5.1 – 10 × ULN | > 10 × ULN |
| M. Urinalysis | | | · | |
| M1. Haematuria | Micro only | Gross, no clots | Clots, transfusion < 2 units | Transfusion required |
| M2. Proteinuria (per 24 h) | 300 – 500 mg (tr/1+) | 501 – 1999 mg (2+) | 2 – 5.0 g (3+) nephrotic syndrome | 5.0 g (4+) anasarca |
| M3. WBC in urine | NA | NA | Indicating acute interstitial nephritis | Associated with acute renal failure |
| M4. Uric acid crystals | Present without symptoms | NA | With stones or symptoms of stones (e.g., renal colic) | Causing renal outflow obstruction and hospitalization |

<sup>\*</sup> In L11,  $1.5 - 1.8 \times ULN$  is changed to  $1.4 - 1.8 \times ULN$ .

<sup>\*\*</sup> In L14,  $1.1 - 2.0 \times ULN$  is changed to  $1.1 - 1.5 \times ULN$ .

<sup>\*\*\*</sup> In L3, L7 and L8, mg/dl is changed to mmol/l.

<sup>\*\*\*\*</sup> For CPK and Creatinine NCI CTC grading will be used. For CPK therefore the following gradings apply: Grade 1: > ULN - 2.5 × ULN; Grade 2: > 2.5 - 5.0 × ULN; Grade 3: > 5.0 - 10.0 × ULN; Grade 4: > 10.0 × ULN; For Creatinine the following gradings apply: Grade 1: > 1 - 1.5 × Baseline; > ULN - 1.5 × ULN; Grade 2: > 1.5 - 3.0 × Baseline; > 1.5 - 3.0 × ULN; Grade 3: > 3.0 baseline; > 3.0 - 6.0 × ULN; Grade 4: > 6.0 × ULN.